CLINICAL TRIAL: NCT04854499
Title: A Phase 2 Study of Magrolimab Combination Therapy in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: Study of Magrolimab Combination Therapy in Patients With Head and Neck Squamous Cell Carcinoma
Acronym: ELEVATE HNSCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-548-5916; 2020-005708-20 (Other: EudraCT Number)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — magrolimab; pembrolizumab; Docetaxel; Fluorouracil; Cisplatin; Carboplatin; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Experimental): Participants with untreated metastatic or unresectable, locally recurrent head and neck squamous cell carcinoma (HNSCC) regardless of programmed cell death ligand 1 (PD-L1) status will receive the following:
  * magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses
  * pembrolizumab 200 mg on Day 1 of each cycle
  * 5-fluorouracil (5-FU) 1000 mg/m^2/day Days 1-4 of each cycle (for up to 6 cycles)
  * platinum chemotherapy (cisplatin 100 mg/m^2 or carboplatin area under the concentration versus time curve (AUC) 5 per investigator choice (for up to 6 cycles)) Participants will continue treatment until unacceptable toxicity or disease progression, whichever occurs first, and will not change their magrolimab dose level after the recommended Phase 2 dose (RP2D) is determined. Each cycle is 21 days.
  Interventions: Drug: Magrolimab; Drug: Pembrolizumab; Drug: 5-FU; Drug: Cisplatin; Drug: Carboplatin
- Safety Run-in Cohort 2, Magrolimab + Docetaxel (Experimental): Participants with locally advanced/metastatic HNSCC regardless of PD-L1 status who were previously treated with at least 1 and no more than 2 lines of prior systemic therapy will receive the following:
  * magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses
  * docetaxel 75 mg/m^2 on Day 1 of each cycle Participants will continue treatment until unacceptable toxicity or disease progression, whichever occurs first, and will not change their magrolimab dose level after the RP2D is determined. Each cycle is 21 days.
  Interventions: Drug: Magrolimab; Drug: Docetaxel
- Pre-expansion Safety Run-in Cohort, Magrolimab + Pembrolizumab (Experimental): The pre-expansion safety run-in cohort may be conducted at the sponsor's discretion prior to the initiation of Phase 2 Cohort 2. Participants with untreated metastatic or unresectable, locally recurrent HNSCC with a PD-L1 combined positive score (CPS) ≥ 1 will receive magrolimab and pembrolizumab 200 mg on Day 1 of each cycle. Each cycle is 21 days.
  Participants will continue treatment until unacceptable toxicity or disease progression, whichever occurs first, and will not change their magrolimab dose level after the RP2D is determined. Each cycle is 21 days.
  Interventions: Drug: Magrolimab; Drug: Pembrolizumab
- Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A) (Experimental): Participants with untreated metastatic or unresectable, locally recurrent HNSCC regardless of PD-L1 status will receive magrolimab at the recommended Phase 2 dose (RP2D) determined in the Safety run-in cohort
  1, pembrolizumab 200 mg on Day 1 of each cycle, 5-FU 1000 mg/m^2/day Days 1-4 of each cycle, and platinum chemotherapy (cisplatin 100 mg/m^2 or carboplatin AUC 5 per investigator choice). Each cycle is 21 days. Magrolimab will be continued until loss of clinical benefit, unacceptable toxicity, or death.
  Pembrolizumab therapy will be administered for up to 24 months or until loss of clinical benefit or unacceptable toxicity, whichever occurs first. 5-FU and platinum chemotherapy will be administered for up to 6 cycles or until loss of clinical benefit or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Magrolimab; Drug: Pembrolizumab; Drug: 5-FU; Drug: Cisplatin; Drug: Carboplatin
- Phase 2 Cohort 1, Pembrolizumab + 5-FU + Platinum (Arm B) (Active Comparator): Participants with untreated metastatic or unresectable, locally recurrent HNSCC regardless of PD-L1 status will receive pembrolizumab 200 mg on Day 1 of each cycle, 5-FU 1000 mg/m^2/day Days 1-4 of each cycle, and platinum chemotherapy (cisplatin 100 mg/m^2 or carboplatin AUC 5 per investigator choice). Each cycle is 21 days.
  Pembrolizumab therapy will be administered for up to 24 months or until loss of clinical benefit or unacceptable toxicity, whichever occurs first. 5-FU and platinum chemotherapy will be administered for up to 6 cycles or until loss of clinical benefit or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: 5-FU; Drug: Cisplatin; Drug: Carboplatin
- Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C) (Active Comparator): Participants with untreated metastatic or unresectable, locally recurrent HNSCC regardless of PD-L1 status will receive magrolimab at the recommended Phase 2 dose (RP2D) determined in the Safety run-in cohort 1, zimberelimab 360 mg on Day 1 of each cycle, 5- FU 1000 mg/m^2/day Days 1-4 of each cycle, and platinum chemotherapy (cisplatin 100 mg/m^2 or carboplatin AUC 5 per investigator choice). Each cycle is 21 days.
  Magrolimab will be continued until loss of clinical benefit, unacceptable toxicity, or death. Zimberelimab therapy will be administered up to 24 months or until loss of clinical benefit or unacceptable toxicity, whichever occurs first. 5-FU and platinum chemotherapy will be administered for up to 6 cycles or until loss of clinical benefit or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Magrolimab; Drug: 5-FU; Drug: Cisplatin; Drug: Carboplatin; Drug: Zimberelimab
- Phase 2 Cohort 2, Magrolimab + Pembrolizumab (Experimental): Participants with untreated metastatic or unresectable, locally recurrent HNSCC with a PD-L1 combined positive score (CPS) ≥ 1 will receive magrolimab at the RP2D determined in the Safety run-in cohort 1 and pembrolizumab 200 mg on Day 1 of each cycle. Each cycle is 21 days.
  Magrolimab will be continued until loss of clinical benefit, unacceptable toxicity, or death. Pembrolizumab therapy will be administered for up to 24 months or until loss of clinical benefit or unacceptable toxicity, whichever occurs first.
  Interventions: Drug: Magrolimab; Drug: Pembrolizumab
- Phase 2 Cohort 3, Magrolimab + Docetaxel (Experimental): Participants with locally advanced/metastatic HNSCC regardless of PD-L1 status who were previously treated with at least 1 and no more than 2 lines of prior systemic therapy will receive magrolimab at the RP2D determined in the Safety run-in cohort 2 and docetaxel 75 mg/m^2 on Day 1 of each cycle. Each cycle is 21 days.
  Magrolimab and docetaxel will be continued until loss of clinical benefit, unacceptable toxicity, or death.
  Interventions: Drug: Magrolimab; Drug: Docetaxel

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: GS-4721
  Arms: Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A); Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C); Phase 2 Cohort 2, Magrolimab + Pembrolizumab; Phase 2 Cohort 3, Magrolimab + Docetaxel; Pre-expansion Safety Run-in Cohort, Magrolimab + Pembrolizumab; Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum; Safety Run-in Cohort 2, Magrolimab + Docetaxel
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
  Arms: Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A); Phase 2 Cohort 2, Magrolimab + Pembrolizumab; Pre-expansion Safety Run-in Cohort, Magrolimab + Pembrolizumab; Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum
Drug: Docetaxel — Administered intravenously
  Arms: Phase 2 Cohort 3, Magrolimab + Docetaxel; Safety Run-in Cohort 2, Magrolimab + Docetaxel
Drug: 5-FU — Administered intravenously
  Arms: Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A); Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C); Phase 2 Cohort 1, Pembrolizumab + 5-FU + Platinum (Arm B); Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum
Drug: Cisplatin — Administered intravenously
  Arms: Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A); Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C); Phase 2 Cohort 1, Pembrolizumab + 5-FU + Platinum (Arm B); Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum
Drug: Carboplatin — Administered intravenously
  Arms: Phase 2 Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum (Arm A); Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C); Phase 2 Cohort 1, Pembrolizumab + 5-FU + Platinum (Arm B); Safety Run-in Cohort 1, Magrolimab + Pembrolizumab + 5-FU + Platinum
Drug: Zimberelimab — Administered intravenously
  Arms: Phase 2 Cohort 1, Magrolimab + Zimberelimab + 5-FU + Platinum (Arm C)

SUMMARY:
The goals of this clinical study are to learn about the safety, tolerability, dosing and effectiveness of the study drug, magrolimab in combination with other anticancer therapies in participants with head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or locally recurrent HNSCC that is considered incurable by local therapies.

Safety Run-in Cohort 1 and Phase 2 Cohorts 1

* Should not have had prior systemic therapy administered in the recurrent or metastatic setting.
* Eligible primary tumor locations include oropharynx, oral cavity, hypopharynx, and larynx. Nasopharynx is not included.
* HNSCC per protocol specified inclusion criteria regardless of PD-L1 status.

Safety Run-in Cohort 2 and Phase 2 Cohort 3

* Histologically or cytologically confirmed locally advanced/mHNSCC regardless of PD-L1 status with at least 1 and no more than 2 lines of prior systemic anticancer therapy in the locally advanced/metastatic setting.

Key Exclusion Criteria:

* Active central nervous system (CNS) disease (individuals with asymptomatic and stable, treated CNS lesions who have been off corticosteroids, radiation, or other CNS-directed therapy for at least 4 weeks are not considered active).
* History of (noninfectious) pneumonitis that required steroids or current pneumonitis.
* Progressive disease within 6 months of completion of curatively intended treatment for locally advanced/mHNSCC.

Safety Run-in Cohort 1, Pre-expansion Safety Run-in Cohort for Magrolimab + Pembrolizumab (if Applicable), and Phase 2 Cohorts 1 and 2

* Prior treatment with any of the following:

  * Anti-programmed cell death protein 1 or anti-PD-L1 checkpoint inhibitors.
  * Anti-cytotoxic T-lymphocyte-associated protein 4 checkpoint inhibitors.

Safety Run-in Cohort 2 and Phase 2 Cohort 3

* Prior treatment with a taxane.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (88):
- United States (22):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - City of Hope, Duarte, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Torrance Memorial Physician Network - Cancer Care Associates, Redondo Beach, California
  - Providence Medical Foundation, Santa Rosa, California
  - Memorial Healthcare System, Hollywood, Florida
  - Ocala Oncology Center, Ocala, Florida
  - University Center and Blood Center,LLC., Athens, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Virginia Piper Cancer Center (Alliant Health, Minneapolis, Minnesota
  - Washington University of Medicine- Siteman Cancer Center, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai and the Mount Sinai Hospital, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (8):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Blacktown Hospital, Westmead, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
- Belgium (7):
  - ZiekenhuisNetwerk Antwerpen (ZNA) - Stuivenberg, Antwerp
  - Algemeen Ziekenhuis Klina, Brasschaat
  - UZ Antwerpen, Edegem
  - Universitaire Ziekenhuis Leuven, Leuven
  - Centre Hospitalizer De L'Ardenne, Libramont-Chevigny
  - AZ Sint-Maarten, Mechelen
  - CHU UCL Namur - Sainte-Elisabeth, Namur
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Centre de Lutte Contre le Cancer (CLCC) - Centre Antoine Lacassagne (CAL) - Site Est, Nice
  - Institut Curie, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Civils de Lyon-Centre Hopitalier Lyon Sud, Pierre-Bénite
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Charite University Medicine, Berlin
  - UniversitÃ¤tsklinikum Bonn, Medizinische Klinik und Poliklinik III, Bonn
  - Universitatsmedizin Gottingen, GÃttingen
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Universitäres Krebszentrum Leipzig, Leipzig
  - Technische Universitat Munchen (TUM) - Klinikum Rechts der Isar, Munich
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Lai Chi Kok
- Italy (7):
  - Azienda Ospedaliero - Universitaria di Bologna - IRCCS, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Ospedale San Luca Luca, Lucca
  - Fondazione IRCCS Istituto Nazionale Tumori Milano, Milan
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico, Modena
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Ospedaliero - Universitaria Senese, Siena
- Poland (5):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Panstwowy Instytut Badawczy, Oddzial x Gliwicach, Gliwice
  - Wielkopolskie Centrum Onkologii im. Marii Sklodowskiej-Curie, Oddzial Onkologii Klinicznej i Immunookologii z Poddoddzialem Dziennym i Izba Przyjec, Poznan
  - Wojewodzki Szpital Specjalistyczny w Siedlcach, Siedlce
  - Narodowy Instytut Onkologii im. M. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Klinika Nowotworow Glowy i Szyi, Warsaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Algarve, Faro
  - Hospital CUF Descobertas, Lisbon
  - Unidade Local de Saude de Matosinhos EPE - Hospital Pedro Hispano SA, Matosinhos Municipality
  - Centro Hospitalar Universitario do Porto, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil,E.P.E., Porto
- Spain (13):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, Royal Marsden - Sutton, London
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colevas AD, Dinis J, Chin V, Costa DA, Park JJ, Fang B, et al. A Phase 2 Study of Magrolimab Combination Therapy in Patients with Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma (ELEVATE HNSCC) [Poster TPS6102]. American Society for Clinical Oncology (ASCO); 2023 June 2-6; Chicago, IL.
- [Background] Colevas AD, Dinis J, Chin V, Costa DA, Park JJ, Fang B, et al. A phase 2 study of magrolimab combination therapy in patients with recurrent or metastatic head and neck squamous cell carcinoma (ELEVATE HNSCC) [Abstract]. American Society for Clinical Oncology (ASCO); 2023 June 2-6; Chicago, IL.
- [Background] Colevas AD, Kerrigan K, Chin V, Rainey N, Park J, Fang B, et al. Safety and Tolerability of Magrolimab Combination Therapy in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (RM-HNSCC) [Poster #675]. SITC: 38th Society for Immunotherapy of Cancer Annual Meeting; 2023 November 3-5, 2023; San Diego, CA.
- [Background] Colevas AD, Kerrigan K, Chin V, Rainey N, Park J, Fang B, et al. Safety and tolerability of magrolimab combination therapy in patients with recurrent or metastatic head and neck squamous cell carcinoma (RM-HNSCC) [Abstract]. SITC: 38th Society for Immunotherapy of Cancer Annual Meeting; 2023 November 3-5, 2023; San Diego, CA.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-548-5916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 279 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in Europe, North America and Asia Pacific. Optional Phase 2 Cohort 2 was never opened due to closure of the study.
Groups:
- Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU: Participants received magrolimab + pembrolizumab + platinum + 5 FU (5-fluorouracil) intravenous (IV) infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 73 weeks; Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 73 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 19 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 18.3 weeks (for carboplatin).
- Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU: Participants received magrolimab + pembrolizumab + platinum + 5 FU IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 72 weeks; Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 88 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 22 weeks for carboplatin and 23 weeks for cisplatin.
- Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU: Participants received pembrolizumab + platinum + 5 FU IV infusions as mentioned below:
  Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 70 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks for carboplatin and 18 weeks for cisplatin.
- Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU: Participants received magrolimab + zimberelimab + platinum + 5 FU IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 37 weeks; Zimberelimab 360 mg IV on Day 1 of every 21-day cycle for up to 40 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 19 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 18 weeks for carboplatin and 16 weeks for cisplatin.
- Safety Run-in Cohort 2: Magrolimab + Docetaxel: Participants received magrolimab + docetaxel IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 69 weeks; Docetaxel 75 mg/m^2 IV on Day 1 of every 21-day cycle for up to 13 weeks.
- Phase 2 Cohort 3: Magrolimab + Docetaxel: Participants received magrolimab + docetaxel IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 42 weeks; Docetaxel 75 mg/m^2 IV on Day 1 of every 21-day cycle for up to 34 weeks.
Period: Overall Study
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel | Phase 2 Cohort 3: Magrolimab + Docetaxel
Started | 6 | 52 | 54 | 32 | 8 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 52 | 54 | 32 | 8 | 41
Not completed — Study Terminated by Sponsor | 5 | 27 | 28 | 19 | 1 | 10
Not completed — Death | 1 | 23 | 21 | 7 | 6 | 24
Not completed — Investigator's Discretion | 0 | 1 | 3 | 4 | 1 | 5
Not completed — Withdrew Consent | 0 | 1 | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Run-in Cohort 1, Safety Run-in Cohort 2 + Phase 2 Cohort 3: The Modified Intent-to-Treat (mITT) Analysis Set included all participants who took at least 1 dose of study drug. Phase 2 Cohort 1: Intent-to-treat (ITT) Analysis Set for Phase 2 Cohort 1 included all participants who were randomized in Phase 2 Cohort 1 of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel | Phase 2 Cohort 3: Magrolimab + Docetaxel | Total
Number analyzed (Participants) | 6 | 52 | 54 | 32 | 7 | 41 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 35 | 33 | 16 | 5 | 22 | 112
  >=65 years | 5 | 17 | 21 | 16 | 2 | 19 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6.2) | 61 (7.4) | 61 (9.5) | 63 (11.4) | 58 (15.5) | 63 (9.9) | 62 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 11 | 5 | 0 | 4 | 29
  Male | 6 | 43 | 43 | 27 | 7 | 37 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 3 | 1 | 1 | 7
  Not Hispanic or Latino | 6 | 43 | 44 | 22 | 6 | 32 | 153
  Unknown or Not Reported | 0 | 7 | 10 | 7 | 0 | 8 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 44 | 47 | 26 | 6 | 30 | 158
  More than one race | 0 | 2 | 1 | 1 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 6 | 5 | 5 | 0 | 7 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 3 | 5 | 1 | 0 | 6 | 15
  United States | 5 | 7 | 8 | 6 | 5 | 11 | 42
  Poland | 0 | 9 | 12 | 7 | 0 | 1 | 29
  Italy | 0 | 1 | 0 | 0 | 0 | 1 | 2
  United Kingdom | 0 | 3 | 0 | 2 | 0 | 0 | 5
  Australia | 1 | 2 | 7 | 3 | 2 | 4 | 19
  France | 0 | 7 | 8 | 9 | 0 | 10 | 34
  Portugal | 0 | 15 | 10 | 1 | 0 | 1 | 27
  Germany | 0 | 0 | 2 | 2 | 0 | 3 | 7
  Spain | 0 | 5 | 2 | 1 | 0 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in Cohorts 1 and 2: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Description: A DLT was defined as any Grade 3 or higher hematologic toxicity or Grade 3 or higher nonhematologic toxicity that had worsened in severity from pretreatment baseline during the DLT assessment period and, in the opinion of the investigator, the AE was related to magrolimab and the relationship of the AE with the combination partner regimen can be ruled out.
Time Frame: First dose date up to 21 days
Population: DLT Evaluable Analysis Set was defined as all participants in the safety run-in evaluations who meet either of the following criteria during the DLT assessment period: The participants experienced a DLT at any time after initiation of the first infusion of magrolimab. The participant didn't experience a DLT and completed at least 2 infusions of magrolimab and at least 1 dose of pembrolizumab, platinum, and 5-FU for Safety Run-in Cohort 1; at least 1 dose of docetaxel for Safety Run-in Cohort 2.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

2. Primary Outcome: Safety Run-in Cohorts 1 and 2: Percentage of Participants Experiencing Grade 3 or 4 Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point up to and including last dose date of study drug plus 30 days (or last dose date of zimberelimab plus 90 days) and prior to the day of initiation of subsequent anti-cancer therapy.
Time Frame: First dose date up to 73 weeks plus 30 days
Population: Safety Run-in Cohorts 1 and 2: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel
Number analyzed (Participants) | 6 | 7
percentage of participants | 83.3 | 71.4

3. Primary Outcome: Phase 2 Cohort 1, Arms A and B: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the earliest date of documented disease progression, as assessed by investigator assessment, or death from any cause, whichever occurred first. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 1, Arms A and B in the ITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum+5-FU: Participants received magrolimab + pembrolizumab + platinum + 5 FU IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 72 weeks; Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 88 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 22 weeks for carboplatin and 23 weeks for cisplatin.
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum+5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU
Number analyzed (Participants) | 52 | 54
months | 5.5 [3.0 to 6.9] | 5.6 [4.2 to 7.4]
Statistical Analysis 1: Comparison: Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum+5-FU vs Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU; Test type: Superiority; Hazard Ratio (HR) = 1.314, 95% CI 2-sided [0.809 to 2.136] — HR along with its 2-sided 95% confidence interval (CI) were estimated using the Cox proportional hazards regression model stratified by the stratification factors at randomization

4. Primary Outcome: Phase 2 Cohort 3: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) as measured by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 as determined by investigator assessment. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 3 in the mITT Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 41
percentage of participants | 12.2 [4.1 to 26.2]

5. Secondary Outcome: Safety Run-in Cohort 1 and 2, Phase 2 Cohort 1 Arm A and Phase 2 Cohort 3: Serum Concentration of Magrolimab
Time Frame: Day 8 1-Hour Postdose; Days 15, 22, 43: Predose; Day 43 1-Hour Postdose; Day 71 1-Hour Postdose; Days 85,127, 190,197, 211, 253 Predose; Day 253 1-Hour Postdose
Population: Participants in the Pharmacokinetic (PK) Analysis Set with available data were analyzed. The PK Analysis Set, defined as all participants who received any amount of magrolimab and have at least 1 evaluable post-treatment serum concentration of magrolimab, at the given timepoint were analyzed. Per pre-specified plan, the PK analysis set included participants from Safety Run-in Cohort 1 and 2, Phase 2 Cohort 1 Arm A and Phase 2 Cohort 3.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 6 | 41 | 6 | 29
μg/mL
  Day 8 1-Hour Postdose: number analyzed (Participants) | 5 | 15 | 5 | 5
  Day 8 1-Hour Postdose | 305 (56.4) | 481 (137) | 288 (55.2) | 459 (140)
  Day 15 Predose: number analyzed (Participants) | 0 | 24 | 0 | 16
  Day 15 Predose |  | 149 (52.8) |  | 125 (49.4)
  Day 22 Predose | 208 (185) | 250 (100) | 255 (149) | 253 (110)
  Day 43 Predose: number analyzed (Participants) | 5 | 38 | 5 | 27
  Day 43 Predose | 359 (253) | 397 (195) | 561 (514) | 477 (219)
  Day 43 1-Hour Postdose: number analyzed (Participants) | 0 | 24 | 0 | 19
  Day 43 1-Hour Postdose |  | 1440 (306) |  | 1330 (426)
  Day 71 1-Hour Postdose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Day 71 1-Hour Postdose |  |  |  | 572 (NA) — Standard Deviation cannot be calculated for one participant.
  Day 85 Predose: number analyzed (Participants) | 4 | 31 | 2 | 18
  Day 85 Predose | 138 (106) | 308 (140) | 813 (830) | 272 (119)
  Day 127 Predose: number analyzed (Participants) | 3 | 4 | 0 | 1
  Day 127 Predose | 142 (113) | 204 (235) |  | 393 (NA) — Standard Deviation cannot be calculated for one participant.
  Day 190 Predose: number analyzed (Participants) | 1 | 12 | 1 | 4
  Day 190 Predose | 707 (NA) — Standard Deviation cannot be calculated for one participant. | 359 (94.9) | NA (0) — Data is not available as the concentrations were below the level of quantification. | 270 (95.9)
  Day 197 Predose: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 197 Predose |  |  | NA (0) — Data is not available as the concentrations were below the level of quantification. |
  Day 211 Predose: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 211 Predose |  | 74.8 (NA) — Standard Deviation cannot be calculated for one participant. |  |
  Day 253 Predose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 253 Predose | 543 (NA) — Standard Deviation cannot be calculated for one participant. | 252 (NA) — Standard Deviation cannot be calculated for one participant. |  |
  Day 253 1-Hour Postdose: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 253 1-Hour Postdose |  | 228 (NA) — Standard Deviation cannot be calculated for one participant. |  |

6. Secondary Outcome: Safety Run-in Cohort 1 and 2, Phase 2 Cohort 1 Arm A, C and Phase 2 Cohort 3: Percentage of Participants Who Developed Antidrug Antibodies (ADAs) to Magrolimab
Time Frame: Up to end of treatment (up to approximately 73 weeks)
Population: Participants in the Immunogenicity Analysis Set with available data were analyzed. The Immunogenicity Analysis Set included all participants who received any amount of magrolimab and have at least 1 evaluable anti-magrolimab antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 6 | 41 | 0 | 32 | 7 | 40
percentage of participants
  ADA Prevalence: number analyzed (Participants) | 6 | 41 | 0 | 0 | 7 | 32
  ADA Prevalence | 16.7 | 3.8 |  |  | 0 | 5.0
  ADA Incidence: number analyzed (Participants) | 6 | 41 | 0 | 32 | 6 | 40
  ADA Incidence | 0 | 0 |  | 3.1 | 0 | 3.1

7. Secondary Outcome: Phase 2 Cohort 1, Arms B and C: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization (Phase 2 Cohorts 1) or date of dose initiation (Phase 2 Cohorts 2 and 3) until the earliest date of documented disease progression as determined by investigator assessment per RECIST, version 1.1, or death from any cause, whichever occurs first. Disease progression is defined in OM#2. KM estimates were used in outcome measure analysis.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 1 Arms B and C in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU
Number analyzed (Participants) | 54 | 32
months | 5.6 [4.2 to 7.4] | 5.5 [3.0 to 9.2]
Statistical Analysis 1: Comparison: Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU vs Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU; Test type: Superiority; Hazard Ratio (HR) = 1.094, 95% CI 2-sided [0.603 to 1.985]

8. Secondary Outcome: Phase 2 Cohort 1, Arms A, B and C: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a CR or PR as determined by investigator assessment. CR and PR are defined in OM#3.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 1, Arms A, B and C in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU
Number analyzed (Participants) | 52 | 54 | 32
percentage of participants | 38.5 [25.3 to 53.0] | 38.9 [25.9 to 53.1] | 37.5 [21.1 to 56.3]
Statistical Analysis 1: Comparison: Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU vs Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU; Test type: Other; Odds Ratio (OR) = 0.982, 95% CI 2-sided [0.449 to 2.147] — The 2-sided 95% CI is based on Clopper-Pearson method
Statistical Analysis 2: Comparison: Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU vs Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU; Test type: Other; Odds Ratio (OR) = 0.943, 95% CI 2-sided [0.383 to 2.321] — The 2-sided 95% CI is based on Clopper-Pearson method

9. Secondary Outcome: Phase 2 Cohort 3: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of dose initiation (Phase 2 Cohort 3) until the earliest date of documented disease progression as determined by investigator assessment per RECIST, version 1.1, or death from any cause, whichever occurs first. Disease progression is defined in OM#2. KM estimates were used in outcome measure analysis
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 3 in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 41
months | 3.6 [2.4 to 4.8]

10. Secondary Outcome: All Phase 2 Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from first documentation of CR or PR to the earliest date of documented disease progression or death from any cause, whichever occurs first. Disease progression is defined in OM#2 and CR and PR are defined in OM#3.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 1, Arms A, B and C in the ITT and participants in Phase 2 Cohort 3 in the mITT analysis set who achieved overall response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 Cohort 1 Arm A: Magrolimab+ Pembrolizumab + Platinum + 5-FU: Participants received magrolimab + pembrolizumab + platinum + 5 FU IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 72 weeks; Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 88 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 22 weeks for carboplatin and 23 weeks for cisplatin.
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab+ Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 20 | 21 | 12 | 5
months | 5.4 [3.5 to 9.3] | 6.2 [3.6 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 6.3 [2.8 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 5.0 [3.3 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

11. Secondary Outcome: All Phase 2 Cohorts: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization (Phase 2 Cohorts 1) or time from the date of dose initiation (Phase 2) to death from any cause. KM estimates were used in outcome measure analysis.
Time Frame: Up to 129 weeks
Population: Participants in Phase 2 Cohort 1, Arms A, B and C in the ITT and participants in Phase 2 Cohort 3 in the mITT analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 52 | 54 | 32 | 41
months | 10.8 [6.9 to 18.2] | 13.3 [9.1 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | NA [7.9 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | 9.1 [6.6 to 12.7]

12. Secondary Outcome: Phase 2 Cohorts: Change From Baseline in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 is a quality of life (QOL) questionnaire for cancer participants, that has 30 items. 5 functional scales (physical, role, emotional, cognitive, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial difficulties). Scoring of the QLQ-C30 was performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the participant), while higher scores on the symptom and single-item scales indicated a higher level of symptoms (i.e. a worse state of the participant).
Time Frame: Baseline, Week 3, Week 6, Week 9, Week 12, Week 15, Week 18, Week 21, Week 24, Week 27 and Week 90
Population: Phase 2 Cohort 1: Participants in the Intent to Treat Analysis Set with available data were analyzed. Phase 2 Cohort 3: Participants in the Modified Intent-to-Treat analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Phase 2 Cohort 1 Arm B: Pembrolizumab+ Platinum+5-FU: Participants received pembrolizumab + platinum + 5 FU IV infusions as mentioned below:
  Pembrolizumab 200 mg IV on Day 1 of every 21-day cycle for up to 70 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 24 weeks for carboplatin and 18 weeks for cisplatin.
- Phase 2 Cohort 3: Magrolimab+Docetaxel: Participants received magrolimab + docetaxel IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 42 weeks; Docetaxel 75 mg/m^2 IV on Day 1 of every 21-day cycle for up to 34 weeks.
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab+ Platinum+5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Phase 2 Cohort 3: Magrolimab+Docetaxel
Number analyzed (Participants) | 52 | 50 | 28 | 37
score on scale
  Global Health Status / QoL: Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Global Health Status / QoL: Baseline | 54.7 (24.9) | 57.3 (23.2) | 55.1 (20.8) | 55.4 (25.6)
  Global Health Status / QoL: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Global Health Status / QoL: Change from Baseline at Week 3 | 5.0 (20.2) | 1.9 (23.3) | -3.6 (16.1) | 1.7 (18.1)
  Global Health Status / QoL: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 26
  Global Health Status / QoL: Change from Baseline at Week 6 | 6.0 (26.5) | 10.2 (26.7) | -1.0 (16.9) | -1.3 (23.7)
  Global Health Status / QoL: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 18 | 21
  Global Health Status / QoL: Change from Baseline at Week 9 | 2.8 (22.2) | 1.1 (27.6) | -4.2 (18.6) | 2.0 (19.0)
  Global Health Status / QoL: Change from Baseline at Week 12: number analyzed (Participants) | 31 | 34 | 17 | 18
  Global Health Status / QoL: Change from Baseline at Week 12 | -4.8 (29.2) | 6.4 (25.8) | 2.9 (14.1) | -4.2 (20.5)
  Global Health Status / QoL: Change from Baseline at Week 15: number analyzed (Participants) | 30 | 29 | 13 | 18
  Global Health Status / QoL: Change from Baseline at Week 15 | -0.3 (27.0) | 5.2 (25.8) | 2.6 (22.7) | 0.0 (24.8)
  Global Health Status / QoL: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Global Health Status / QoL: Change from Baseline at Week 18 | 5.4 (27.0) | 10.0 (26.4) | -4.5 (23.1) | -2.8 (23.7)
  Global Health Status / QoL: Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 10 | 13
  Global Health Status / QoL: Change from Baseline at Week 21 | 4.3 (28.1) | 4.9 (22.4) | -10.8 (23.6) | -8.3 (20.7)
  Global Health Status / QoL: Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 12 | 9
  Global Health Status / QoL: Change from Baseline at Week 24 | 9.2 (26.3) | 1.9 (20.9) | -5.6 (23.9) | -10.2 (15.5)
  Global Health Status / QoL: Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 6 | 5
  Global Health Status / QoL: Change from Baseline at Week 27 | 2.2 (27.7) | 0.0 (18.6) | 6.9 (26.0) | 1.7 (24.6)
  Global Health Status / QoL: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Global Health Status / QoL: Change from Baseline at Week 90 | 33.3 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Functional Scales: Physical Functioning: Baseline: number analyzed (Participants) | 52 | 50 | 27 | 37
  Functional Scales: Physical Functioning: Baseline | 75.0 (25.3) | 75.4 (23.2) | 74.9 (23.2) | 73.7 (23.8)
  Functional Scales: Physical Functioning: Change from Baseline at Week 3: number analyzed (Participants) | 43 | 43 | 22 | 29
  Functional Scales: Physical Functioning: Change from Baseline at Week 3 | -4.8 (15.6) | -3.6 (21.2) | -9.2 (15.7) | -2.9 (17.0)
  Functional Scales: Physical Functioning: Change from Baseline at Week 6: number analyzed (Participants) | 33 | 36 | 15 | 27
  Functional Scales: Physical Functioning: Change from Baseline at Week 6 | -3.4 (14.4) | 2.2 (20.2) | -6.2 (15.6) | -11.3 (21.7)
  Functional Scales: Physical Functioning: Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 18 | 21
  Functional Scales: Physical Functioning: Change from Baseline at Week 9 | -1.4 (21.3) | -1.0 (18.8) | -4.3 (15.9) | -2.9 (13.9)
  Functional Scales: Physical Functioning: Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 16 | 18
  Functional Scales: Physical Functioning: Change from Baseline at Week 12 | -4.5 (22.7) | 3.8 (23.7) | -5.3 (15.7) | -10.0 (17.5)
  Functional Scales: Physical Functioning: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 12 | 18
  Functional Scales: Physical Functioning: Change from Baseline at Week 15 | -6.5 (21.0) | 3.3 (26.2) | -13.3 (24.1) | -11.9 (19.7)
  Functional Scales: Physical Functioning: Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 10 | 15
  Functional Scales: Physical Functioning: Change from Baseline at Week 18 | 0.0 (15.5) | 2.7 (27.7) | -4.7 (13.4) | -16.0 (20.7)
  Functional Scales: Physical Functioning: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Functional Scales: Physical Functioning: Change from Baseline at Week 21 | -5.0 (20.9) | -6.5 (21.4) | -12.1 (19.3) | -21.0 (24.2)
  Functional Scales: Physical Functioning: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 12 | 9
  Functional Scales: Physical Functioning: Change from Baseline at Week 24 | -5.1 (15.9) | -7.4 (23.6) | -8.3 (14.0) | -21.5 (10.9)
  Functional Scales: Physical Functioning: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Functional Scales: Physical Functioning: Change from Baseline at Week 27 | -7.9 (17.6) | 0.0 (20.3) | -12.0 (14.5) | -22.7 (18.0)
  Functional Scales: Physical Functioning: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Functional Scales: Physical Functioning: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Functional Scales: Role Functioning: Baseline: number analyzed (Participants) | 52 | 49 | 27 | 37
  Functional Scales: Role Functioning: Baseline | 72.8 (32.5) | 74.5 (27.7) | 69.8 (32.0) | 60.8 (35.4)
  Functional Scales: Role Functioning: Change from Baseline at Week 3: number analyzed (Participants) | 43 | 41 | 22 | 29
  Functional Scales: Role Functioning: Change from Baseline at Week 3 | -1.9 (21.6) | -2.4 (33.9) | -12.1 (37.2) | -5.7 (28.3)
  Functional Scales: Role Functioning: Change from Baseline at Week 6: number analyzed (Participants) | 33 | 35 | 15 | 26
  Functional Scales: Role Functioning: Change from Baseline at Week 6 | -5.1 (23.4) | 2.4 (32.6) | -10.0 (19.7) | -3.2 (26.7)
  Functional Scales: Role Functioning: Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 18 | 9
  Functional Scales: Role Functioning: Change from Baseline at Week 9 | -3.6 (29.2) | -5.6 (35.1) | -9.3 (30.4) | 7.9 (27.2)
  Functional Scales: Role Functioning: Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 16 | 18
  Functional Scales: Role Functioning: Change from Baseline at Week 12 | -6.2 (35.9) | 2.0 (38.0) | -7.3 (33.3) | -8.3 (37.6)
  Functional Scales: Role Functioning: Change from Baseline at Week 15: number analyzed (Participants) | 32 | 29 | 12 | 18
  Functional Scales: Role Functioning: Change from Baseline at Week 15 | -10.4 (36.4) | 7.5 (35.8) | -6.9 (28.8) | -4.6 (32.2)
  Functional Scales: Role Functioning: Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 10 | 15
  Functional Scales: Role Functioning: Change from Baseline at Week 18 | -4.0 (30.7) | -1.3 (37.1) | -5.0 (19.3) | -7.8 (37.2)
  Functional Scales: Role Functioning: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 23 | 11 | 13
  Functional Scales: Role Functioning: Change from Baseline at Week 21 | -6.9 (38.0) | -11.6 (29.1) | -13.6 (35.6) | -14.1 (39.0)
  Functional Scales: Role Functioning: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 12 | 9
  Functional Scales: Role Functioning: Change from Baseline at Week 24 | -4.8 (32.6) | -2.8 (30.9) | 0.0 (24.6) | -20.4 (21.7)
  Functional Scales: Role Functioning: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Functional Scales: Role Functioning: Change from Baseline at Week 27 | -16.7 (21.1) | -11.1 (37.1) | -10.0 (22.4) | -23.3 (19.0)
  Functional Scales: Role Functioning: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Functional Scales: Role Functioning: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Functional Scales: Emotional Functioning: Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Functional Scales: Emotional Functioning: Baseline | 69.5 (25.3) | 69.7 (27.6) | 70.3 (28.3) | 81.5 (16.4)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Functional Scales: Emotional Functioning: Change from Baseline at Week 3 | 7.7 (25.1) | 7.5 (25.2) | 5.7 (20.9) | 1.2 (17.5)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 26
  Functional Scales: Emotional Functioning: Change from Baseline at Week 6 | 12.6 (23.5) | 12.3 (25.9) | 4.0 (24.6) | -5.7 (21.8)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 18 | 21
  Functional Scales: Emotional Functioning: Change from Baseline at Week 9 | 7.7 (19.8) | 6.1 (16.5) | 11.4 (22.6) | 0.1 (14.8)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 12: number analyzed (Participants) | 31 | 34 | 17 | 18
  Functional Scales: Emotional Functioning: Change from Baseline at Week 12 | 3.8 (24.6) | 11.8 (20.7) | 9.6 (21.0) | 1.5 (11.6)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 15: number analyzed (Participants) | 30 | 29 | 13 | 18
  Functional Scales: Emotional Functioning: Change from Baseline at Week 15 | 0.3 (28.0) | 11.8 (27.1) | 3.6 (19.8) | -5.4 (19.3)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Functional Scales: Emotional Functioning: Change from Baseline at Week 18 | 3.7 (23.8) | 12.0 (25.8) | 6.6 (28.6) | -4.4 (16.5)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 10 | 13
  Functional Scales: Emotional Functioning: Change from Baseline at Week 21 | 0.8 (22.6) | 2.0 (22.5) | 6.7 (12.3) | -5.6 (12.7)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 13 | 9
  Functional Scales: Emotional Functioning: Change from Baseline at Week 24 | 3.1 (20.0) | 4.6 (22.4) | 2.4 (19.8) | -4.3 (9.0)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 6 | 5
  Functional Scales: Emotional Functioning: Change from Baseline at Week 27 | 0.6 (16.5) | 9.6 (10.9) | 6.5 (27.6) | -11.1 (18.1)
  Functional Scales: Emotional Functioning: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Functional Scales: Emotional Functioning: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Functional Scales : Cognitive Functioning : Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Functional Scales : Cognitive Functioning : Baseline | 84.0 (22.1) | 84.7 (22.3) | 85.7 (16.8) | 83.8 (21.3)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 3 | 1.6 (16.0) | -0.4 (20.7) | -7.2 (14.1) | -4.6 (16.6)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 26
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 6 | 2.1 (15.7) | 0.9 (25.8) | -1.0 (7.4) | -2.6 (24.4)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 18 | 21
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 9 | 1.9 (14.1) | -0.6 (14.8) | -2.8 (13.1) | -4.8 (19.1)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 12: number analyzed (Participants) | 31 | 34 | 17 | 18
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 12 | -6.5 (23.8) | 1.5 (18.5) | -4.9 (12.9) | -3.7 (20.3)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 15 | -3.8 (22.2) | 0.6 (19.1) | -1.3 (12.7) | -1.9 (13.9)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 18 | -4.8 (22.2) | -1.3 (20.9) | -6.1 (8.4) | -3.3 (16.9)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 10 | 13
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 21 | -3.6 (20.1) | -0.7 (18.7) | -6.7 (8.6) | -10.3 (26.8)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 13 | 9
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 24 | -3.3 (16.8) | -3.7 (18.6) | -3.8 (12.1) | -13.0 (16.2)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 6 | 5
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 27 | 0.0 (15.4) | -4.4 (11.7) | -5.6 (8.6) | -33.3 (31.2)
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Functional Scales : Cognitive Functioning : Change from Baseline at Week 90 | 16.7 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Functional Scales : Social Functioning : Baseline: number analyzed (Participants) | 51 | 49 | 28 | 37
  Functional Scales : Social Functioning : Baseline | 75.5 (26.5) | 73.8 (31.2) | 76.8 (24.1) | 68.0 (36.9)
  Functional Scales : Social Functioning : Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Functional Scales : Social Functioning : Change from Baseline at Week 3 | 2.4 (24.6) | -3.5 (33.6) | -12.3 (23.7) | -3.4 (30.3)
  Functional Scales : Social Functioning : Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 26
  Functional Scales : Social Functioning : Change from Baseline at Week 6 | 3.6 (27.7) | 6.9 (33.4) | -7.3 (18.2) | 1.3 (35.6)
  Functional Scales : Social Functioning : Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 18 | 21
  Functional Scales : Social Functioning : Change from Baseline at Week 9 | -3.7 (28.6) | -3.3 (23.3) | -7.4 (21.6) | 9.5 (34.0)
  Functional Scales : Social Functioning : Change from Baseline at Week 12: number analyzed (Participants) | 31 | 33 | 17 | 18
  Functional Scales : Social Functioning : Change from Baseline at Week 12 | -2.2 (30.0) | 0.5 (31.0) | -4.9 (19.3) | -7.4 (27.5)
  Functional Scales : Social Functioning : Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Functional Scales : Social Functioning : Change from Baseline at Week 15 | -8.1 (34.1) | 4.0 (27.7) | 5.1 (23.0) | -2.8 (41.3)
  Functional Scales : Social Functioning : Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Functional Scales : Social Functioning : Change from Baseline at Week 18 | 1.2 (22.6) | 2.7 (19.6) | -1.5 (15.7) | 7.8 (36.1)
  Functional Scales : Social Functioning : Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 10 | 13
  Functional Scales : Social Functioning : Change from Baseline at Week 21 | -5.8 (30.0) | -0.7 (24.3) | -11.7 (28.4) | -5.1 (41.6)
  Functional Scales : Social Functioning : Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 13 | 9
  Functional Scales : Social Functioning : Change from Baseline at Week 24 | -0.8 (28.9) | -4.6 (32.7) | -1.3 (22.0) | -22.2 (25.0)
  Functional Scales : Social Functioning : Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 6 | 5
  Functional Scales : Social Functioning : Change from Baseline at Week 27 | -2.2 (30.8) | -5.6 (12.1) | -5.6 (13.6) | -33.3 (31.2)
  Functional Scales : Social Functioning : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Functional Scales : Social Functioning : Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Fatigue: Baseline | 37.4 (28.9) | 38.6 (24.3) | 40.1 (30.3) | 42.9 (29.9)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 3: number analyzed (Participants) | 43 | 43 | 23 | 29
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 3 | 1.7 (19.7) | 2.5 (20.8) | 7.2 (26.7) | 8.0 (25.7)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 6: number analyzed (Participants) | 33 | 36 | 16 | 27
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 6 | -2.7 (21.9) | -5.4 (27.3) | 4.2 (27.5) | 13.2 (28.9)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 19 | 21
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 9 | 0.4 (22.5) | -0.2 (31.2) | 3.8 (29.5) | -3.2 (26.8)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 17 | 37
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 12 | 2.8 (24.1) | -4.4 (26.9) | 2.0 (26.1) | 8.6 (27.5)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 15 | 8.6 (28.4) | -4.4 (27.5) | 8.5 (36.6) | 12.3 (24.7)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 11 | 15
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 18 | 4.2 (23.8) | -2.6 (25.5) | 7.1 (36.6) | 18.5 (31.6)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 21 | 3.7 (27.3) | 2.5 (23.9) | 11.6 (40.2) | 15.4 (30.6)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 24 | 4.8 (22.4) | 0.9 (24.9) | 7.7 (29.9) | 29.6 (15.7)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 27 | 2.1 (17.8) | 4.8 (27.8) | 2.2 (25.3) | 35.6 (24.1)
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Fatigue: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Nausea and Vomiting : Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Symptom Scales / Items: Nausea and Vomiting : Baseline | 5.6 (16.6) | 5.7 (12.4) | 4.8 (11.9) | 7.7 (15.5)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 3 | 6.7 (20.2) | 5.0 (16.5) | 15.9 (34.3) | 2.9 (12.7)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 6: number analyzed (Participants) | 33 | 36 | 16 | 27
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 6 | 1.0 (13.8) | 2.3 (21.1) | 2.1 (16.0) | 0.6 (16.3)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 19 | 21
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 9 | 8.6 (25.1) | 3.9 (20.4) | 7.9 (25.1) | 5.6 (21.3)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 12: number analyzed (Participants) | 30 | 34 | 17 | 18
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 12 | 13.3 (27.5) | 3.9 (18.8) | 1.0 (23.9) | -1.9 (13.9)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 15 | 5.9 (21.8) | 5.7 (22.8) | 5.1 (12.5) | 3.7 (18.6)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 15
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 18 | 3.6 (18.9) | 4.5 (21.9) | 3.0 (10.1) | 5.6 (26.5)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 21 | 7.6 (18.4) | 6.3 (21.3) | 11.1 (29.6) | 7.7 (20.0)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 24 | 4.8 (12.0) | 0.0 (9.9) | 5.1 (12.5) | -1.9 (13.0)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 27 | 2.1 (12.0) | 4.4 (13.3) | 13.3 (18.3) | -3.3 (18.3)
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Nausea and Vomiting : Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Pain : Baseline | 37.2 (32.1) | 40.3 (30.9) | 39.9 (31.5) | 36.0 (33.2)
  Symptom Scales / Items: Pain : Change from Baseline at Week 3: number analyzed (Participants) | 43 | 43 | 23 | 29
  Symptom Scales / Items: Pain : Change from Baseline at Week 3 | -5.8 (27.4) | -3.9 (31.0) | -2.9 (25.5) | -5.7 (27.9)
  Symptom Scales / Items: Pain : Change from Baseline at Week 6: number analyzed (Participants) | 33 | 36 | 16 | 27
  Symptom Scales / Items: Pain : Change from Baseline at Week 6 | -12.1 (22.5) | -19.9 (36.0) | -10.4 (22.7) | -3.7 (34.1)
  Symptom Scales / Items: Pain : Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 19 | 21
  Symptom Scales / Items: Pain : Change from Baseline at Week 9 | -7.7 (23.8) | -13.9 (29.1) | -8.8 (28.5) | -13.5 (28.2)
  Symptom Scales / Items: Pain : Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 17 | 18
  Symptom Scales / Items: Pain : Change from Baseline at Week 12 | -4.7 (28.5) | -23.0 (34.6) | -13.7 (24.5) | -3.7 (31.6)
  Symptom Scales / Items: Pain : Change from Baseline at Week 15: number analyzed (Participants) | 32 | 29 | 13 | 18
  Symptom Scales / Items: Pain : Change from Baseline at Week 15 | -2.6 (31.4) | -19.0 (36.4) | 0.0 (30.4) | -4.6 (34.2)
  Symptom Scales / Items: Pain : Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 11 | 15
  Symptom Scales / Items: Pain : Change from Baseline at Week 18 | -8.0 (22.5) | -18.6 (35.4) | 6.1 (15.4) | -2.2 (30.8)
  Symptom Scales / Items: Pain : Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Pain : Change from Baseline at Week 21 | -1.4 (28.6) | -10.4 (31.8) | -1.4 (35.9) | -6.4 (35.7)
  Symptom Scales / Items: Pain : Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Pain : Change from Baseline at Week 24 | -0.8 (22.0) | -12.0 (29.6) | 0.0 (31.2) | 9.3 (16.9)
  Symptom Scales / Items: Pain : Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Symptom Scales / Items: Pain : Change from Baseline at Week 27 | 9.4 (28.5) | -8.9 (39.3) | 8.3 (17.5) | 16.7 (39.1)
  Symptom Scales / Items: Pain : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Pain : Change from Baseline at Week 90 | -16.7 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Dyspnoea : Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Symptom Scales / Items: Dyspnoea : Baseline | 17.0 (25.3) | 15.3 (24.5) | 22.6 (31.5) | 24.3 (32.1)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 3 | 0.8 (20.1) | 2.3 (28.5) | 1.4 (18.7) | 9.2 (23.4)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 6: number analyzed (Participants) | 32 | 35 | 16 | 27
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 6 | 2.1 (20.6) | -1.9 (27.9) | 6.3 (18.1) | 13.6 (34.9)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 19 | 21
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 9 | 0.0 (22.2) | 10.0 (34.1) | -5.3 (20.1) | 11.1 (21.9)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 17 | 18
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 12 | 3.1 (23.0) | 5.9 (32.3) | 3.9 (20.0) | 0.0 (19.8)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 15 | 10.8 (29.0) | 3.4 (32.5) | 5.1 (26.7) | 13.0 (25.9)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 11 | 15
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 18 | 4.6 (21.3) | 7.7 (30.3) | 9.1 (15.6) | 24.4 (29.5)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 21 | 5.6 (21.2) | 16.7 (32.6) | 11.1 (35.8) | 20.5 (29.0)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 24 | 1.6 (22.3) | 5.6 (32.8) | 7.7 (24.2) | 11.1 (28.9)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 27 | 2.1 (14.8) | 4.4 (24.8) | 6.7 (14.9) | 13.3 (38.0)
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Dyspnoea : Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Insomnia : Baseline | 39.1 (27.0) | 34.7 (30.1) | 34.5 (35.7) | 34.2 (33.8)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 3: number analyzed (Participants) | 43 | 43 | 23 | 29
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 3 | -17.8 (26.6) | 0.0 (32.5) | 2.9 (26.4) | -2.3 (23.5)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 6: number analyzed (Participants) | 33 | 36 | 16 | 26
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 6 | -15.2 (31.3) | -11.1 (39.0) | 14.6 (32.1) | 1.3 (31.9)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 19 | 21
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 9 | -11.9 (35.4) | -20.0 (38.8) | -8.8 (21.8) | -9.5 (23.9)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 12: number analyzed (Participants) | 32 | 34 | 17 | 18
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 12 | -15.6 (40.6) | -16.7 (34.1) | -7.8 (30.1) | -3.7 (25.3)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 15 | -11.8 (36.1) | -13.8 (33.9) | -5.1 (23.0) | -7.4 (31.4)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 18: number analyzed (Participants) | 29 | 26 | 11 | 15
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 18 | -11.5 (27.1) | -7.7 (40.3) | -3.0 (37.9) | 6.7 (28.7)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 21 | -2.8 (27.7) | -6.9 (42.8) | -2.8 (17.2) | -2.6 (41.9)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 24 | -4.8 (30.3) | -11.1 (37.9) | -10.3 (34.4) | 11.1 (33.3)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 27 | 0.0 (36.5) | 2.2 (44.5) | 6.7 (27.9) | 13.3 (50.6)
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Insomnia : Change from Baseline at Week 90 | -33.3 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Appetite Loss: Baseline: number analyzed (Participants) | 52 | 50 | 27 | 36
  Symptom Scales / Items: Appetite Loss: Baseline | 29.5 (37.7) | 20.7 (24.2) | 29.6 (31.1) | 32.4 (36.1)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 3: number analyzed (Participants) | 43 | 43 | 22 | 28
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 3 | 6.2 (29.3) | 7.0 (27.8) | 13.6 (33.6) | 2.4 (33.9)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 6: number analyzed (Participants) | 33 | 35 | 16 | 27
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 6 | -5.1 (29.0) | 0.0 (37.0) | -4.2 (16.7) | -3.7 (36.2)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 9: number analyzed (Participants) | 28 | 30 | 18 | 21
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 9 | 3.6 (36.7) | 2.2 (38.1) | 1.9 (37.0) | -4.8 (33.8)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 12: number analyzed (Participants) | 31 | 33 | 16 | 18
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 12 | 5.4 (44.8) | -1.0 (32.8) | -2.1 (22.7) | 7.4 (50.6)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 12 | 17
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 15 | 6.5 (37.9) | 2.3 (36.7) | 8.3 (28.9) | 5.9 (29.4)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 15
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 18 | 1.2 (32.1) | 2.6 (37.6) | 3.0 (37.9) | 0.0 (39.8)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 12 | 13
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 21 | 6.9 (42.8) | 9.7 (39.9) | 13.9 (38.8) | 2.6 (39.6)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 18 | 13 | 9
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 24 | 3.2 (27.7) | 1.9 (33.3) | 5.1 (32.9) | 7.4 (36.4)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 5 | 5
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 27 | 14.6 (34.4) | 4.4 (30.5) | 6.7 (14.9) | 13.3 (38.0)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Constipation: Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Symptom Scales / Items: Constipation: Baseline | 23.5 (30.0) | 27.3 (30.6) | 25.0 (29.6) | 21.6 (28.6)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Symptom Scales / Items: Constipation: Change from Baseline at Week 3 | 0.8 (23.8) | -3.1 (33.2) | 5.8 (32.8) | 2.3 (21.7)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Symptom Scales / Items: Constipation: Change from Baseline at Week 6 | -6.3 (33.3) | -1.9 (33.8) | 0.0 (32.2) | 0.0 (20.7)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 19 | 21
  Symptom Scales / Items: Constipation: Change from Baseline at Week 9 | 3.7 (32.5) | -2.2 (38.1) | -7.0 (23.8) | 1.6 (26.8)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 12: number analyzed (Participants) | 30 | 34 | 17 | 18
  Symptom Scales / Items: Constipation: Change from Baseline at Week 12 | -2.2 (36.0) | -1.0 (32.3) | -2.0 (27.6) | 3.7 (27.7)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 29 | 13 | 18
  Symptom Scales / Items: Constipation: Change from Baseline at Week 15 | -2.2 (31.0) | -2.3 (39.8) | 0.0 (36.0) | 11.1 (36.2)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 15
  Symptom Scales / Items: Constipation: Change from Baseline at Week 18 | -7.1 (31.9) | -3.8 (38.1) | 0.0 (14.9) | 6.7 (31.4)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 12 | 13
  Symptom Scales / Items: Constipation: Change from Baseline at Week 21 | -7.2 (31.7) | 1.4 (39.9) | -8.3 (25.1) | 5.1 (23.0)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 13 | 9
  Symptom Scales / Items: Constipation: Change from Baseline at Week 24 | -10.0 (40.6) | 1.9 (47.8) | -5.1 (23.0) | 0.0 (23.6)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 5 | 5
  Symptom Scales / Items: Constipation: Change from Baseline at Week 27 | -6.7 (42.2) | 4.4 (41.5) | -6.7 (14.9) | 0.0 (23.6)
  Symptom Scales / Items: Constipation: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Constipation: Change from Baseline at Week 90 | -33.3 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Diarrhoea: Baseline: number analyzed (Participants) | 51 | 50 | 28 | 37
  Symptom Scales / Items: Diarrhoea: Baseline | 5.2 (12.2) | 8.7 (20.0) | 2.4 (8.7) | 7.2 (17.8)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 43 | 23 | 29
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 3 | 4.0 (16.8) | 0.8 (21.2) | 10.1 (23.4) | 5.7 (33.4)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 26
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 6 | 0.0 (14.7) | -1.9 (17.7) | 4.2 (11.4) | 3.8 (35.7)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 30 | 18 | 21
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 9 | 6.2 (26.2) | -1.1 (22.3) | 9.3 (25.1) | -1.6 (19.7)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 12: number analyzed (Participants) | 31 | 33 | 17 | 18
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 12 | 4.3 (20.6) | 0.0 (18.6) | 5.9 (13.1) | 7.4 (21.6)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 15: number analyzed (Participants) | 30 | 29 | 13 | 18
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 15 | 8.9 (26.2) | -3.4 (24.1) | 10.3 (21.0) | 11.1 (32.3)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 18 | 0.0 (15.7) | -4.0 (20.0) | 6.1 (13.5) | 11.1 (24.1)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 10 | 13
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 21 | 0.0 (10.1) | 4.2 (22.7) | 6.7 (14.1) | 17.9 (22.0)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 24: number analyzed (Participants) | 20 | 18 | 13 | 9
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 24 | 1.7 (13.1) | -7.4 (18.3) | 10.3 (21.0) | 14.8 (37.7)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 27: number analyzed (Participants) | 15 | 15 | 6 | 5
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 27 | 6.7 (13.8) | -4.4 (27.8) | 11.1 (17.2) | 13.3 (38.0)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |
  Symptom Scales / Items: Financial Difficulties: Baseline: number analyzed (Participants) | 51 | 48 | 28 | 34
  Symptom Scales / Items: Financial Difficulties: Baseline | 16.3 (26.1) | 22.2 (32.5) | 17.9 (29.4) | 14.7 (29.8)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 42 | 23 | 26
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 3 | -2.4 (26.9) | 1.6 (32.9) | 5.8 (21.7) | -2.6 (20.9)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 35 | 16 | 24
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 6 | -2.1 (18.8) | 2.9 (31.7) | 6.3 (25.0) | 1.4 (20.8)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 29 | 18 | 19
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 9 | -1.2 (29.9) | 3.4 (25.7) | -1.9 (13.9) | -7.0 (30.6)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 12: number analyzed (Participants) | 31 | 33 | 17 | 16
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 12 | 3.2 (32.6) | 8.1 (28.9) | 0.0 (16.7) | 6.3 (32.7)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 17
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 15 | 8.9 (30.2) | 1.2 (32.1) | -5.1 (18.5) | 0.0 (23.6)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 24 | 11 | 13
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 18 | 0.0 (24.0) | 2.8 (16.8) | -3.0 (10.1) | -5.1 (35.6)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 21: number analyzed (Participants) | 23 | 23 | 10 | 11
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 21 | 0.0 (22.5) | 0.0 (28.4) | -3.3 (10.5) | -3.0 (31.5)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 7
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 24 | 5.0 (12.2) | 5.9 (21.2) | 0.0 (13.6) | 19.0 (32.5)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 27: number analyzed (Participants) | 15 | 14 | 6 | 4
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 27 | 8.9 (15.3) | 4.8 (17.8) | 0.0 (21.1) | 0.0 (0.0)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Week 90 | 0.0 (NA) — Standard deviation cannot be calculated for one participant. |  |  |

13. Secondary Outcome: Phase 2 Cohorts: Change From Baseline in the European Organisation for Research and Treatment of Cancer Quality of Life - Head and Neck Module (EORTC QLQ-H&N35)
Description: The H&N35 is a 35-item questionnaire for participants with H&N cancer. It includes 7 multi-item scales that assess pain (4 items), swallowing (4 items), senses (2 items), speech (3 items), social eating (4 items), social contact (5 items), and sexuality (2 items). There are also 11 single items: teeth, opening mouth, dry mouth, sticky saliva, coughing, felt ill, pain killers, nutritional supplements, feeding tube, weight loss, weight gain. All symptoms scales, scores were transformed in range of 0 to 100, where higher scores indicated more severe symptoms. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 3, Week 6, Week 9, Week 12, Week 15, Week 18, Week 21, Week 24, Week 27, and Week 90
Population: Phase 2 Cohort 1: Participants in the Intent-to-Treat Analysis Set with available data were analyzed. Phase 2 Cohort 3: Participants in the Modified Intent-to-Treat Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 52 | 49 | 28 | 37
score on scale
  Parameter: Symptom Scales / Items : Pain; Baseline | 27.1 (30.6) | 26.7 (24.8) | 28.7 (25.2) | 25.0 (25.4)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 3: number analyzed (Participants) | 42 | 42 | 23 | 29
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 3 | -2.8 (27.3) | 3.0 (22.8) | 6.0 (15.3) | -5.7 (21.9)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 6 | -4.7 (22.7) | -2.9 (31.8) | 0.0 (23.6) | -4.6 (23.7)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 9: number analyzed (Participants) | 28 | 29 | 19 | 21
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 9 | -2.1 (24.5) | -3.2 (22.4) | 2.3 (33.1) | -6.0 (29.1)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 12: number analyzed (Participants) | 32 | 33 | 17 | 19
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 12 | -5.2 (24.7) | -7.9 (29.1) | -4.6 (26.5) | 3.9 (21.2)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 15: number analyzed (Participants) | 31 | 28 | 13 | 18
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 15 | 2.4 (25.6) | -5.7 (30.6) | -5.8 (24.9) | -7.4 (28.9)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 18 | -2.1 (21.7) | -10.3 (29.1) | 6.8 (16.2) | -1.2 (15.3)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 21 | 2.1 (27.6) | -1.7 (34.6) | -6.8 (19.3) | -4.5 (31.1)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 24 | -3.6 (21.8) | -11.8 (37.6) | -4.5 (15.1) | 2.2 (24.6)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 27 | -4.2 (24.7) | -10.6 (36.1) | -6.9 (24.4) | 5.0 (22.5)
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items : Pain; Change from Baseline at Week 90 | -58.3 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Swallowing; Baseline: number analyzed (Participants) | 51 | 49 | 28 | 36
  Parameter: Symptom Scales / Items: Swallowing; Baseline | 30.1 (33.2) | 33.6 (34.8) | 31.0 (26.1) | 36.3 (31.9)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 40 | 23 | 28
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 3 | -4.3 (24.6) | 2.3 (24.5) | 4.1 (21.3) | -3.4 (20.9)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 6: number analyzed (Participants) | 30 | 35 | 16 | 26
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 6 | -9.7 (22.5) | -8.3 (29.7) | -3.1 (22.1) | -7.7 (24.5)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 9: number analyzed (Participants) | 28 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 9 | -5.9 (24.0) | -6.6 (24.9) | 0.4 (25.5) | -9.0 (31.1)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 12: number analyzed (Participants) | 31 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 12 | -6.9 (25.0) | -3.3 (21.5) | -5.4 (15.9) | -3.5 (20.8)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 15: number analyzed (Participants) | 31 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 15 | -3.0 (29.2) | -0.3 (23.0) | -8.3 (19.2) | -8.3 (23.7)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 18 | -5.1 (28.9) | 0.0 (32.8) | -2.3 (10.6) | -3.6 (15.6)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 21 | -2.2 (25.0) | 5.7 (33.3) | -3.8 (13.6) | -15.0 (29.8)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 24 | -3.3 (23.0) | -1.0 (18.1) | -2.6 (18.4) | 0.0 (20.4)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 27 | 5.7 (22.7) | -5.6 (21.1) | -13.9 (11.4) | -1.7 (12.4)
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Swallowing; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Senses Problems; Baseline: number analyzed (Participants) | 52 | 49 | 28 | 36
  Parameter: Symptom Scales / Items: Senses Problems; Baseline | 16.0 (25.8) | 23.5 (30.6) | 18.5 (26.2) | 29.2 (29.4)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 3: number analyzed (Participants) | 42 | 42 | 23 | 29
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 3 | -0.4 (21.0) | -1.2 (21.3) | 0.7 (19.8) | -4.0 (25.8)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 6 | -4.2 (21.2) | 2.8 (30.5) | 9.4 (14.9) | 1.9 (22.3)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 9: number analyzed (Participants) | 28 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 9 | -3.6 (21.4) | 0.6 (22.9) | 3.5 (28.1) | 0.8 (18.6)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 12: number analyzed (Participants) | 32 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 12 | 2.1 (14.5) | -2.5 (24.3) | -4.9 (28.1) | 3.5 (27.5)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 15: number analyzed (Participants) | 32 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 15 | 1.0 (25.4) | 0.6 (25.0) | -2.6 (16.5) | 3.7 (16.7)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 18 | 4.2 (27.8) | -7.1 (17.1) | -1.5 (11.7) | 6.0 (26.6)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 21 | 3.5 (26.5) | 4.9 (31.3) | 1.5 (13.9) | -1.3 (19.8)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 24 | 2.4 (29.0) | 3.9 (25.4) | -1.3 (12.7) | -3.7 (27.4)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 27 | 8.3 (40.4) | -2.2 (17.7) | -5.6 (13.6) | 13.3 (13.9)
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Senses Problems; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Speech Problems; Baseline: number analyzed (Participants) | 51 | 48 | 28 | 36
  Parameter: Symptom Scales / Items: Speech Problems; Baseline | 36.2 (32.7) | 32.1 (31.0) | 32.1 (27.8) | 29.3 (30.8)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 3: number analyzed (Participants) | 40 | 40 | 23 | 28
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 3 | -6.7 (22.2) | -1.1 (19.9) | 0.5 (19.1) | 4.2 (26.0)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 6: number analyzed (Participants) | 29 | 35 | 16 | 25
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 6 | -11.9 (21.4) | -6.3 (29.6) | -2.1 (20.8) | -1.3 (27.1)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 9: number analyzed (Participants) | 26 | 29 | 19 | 20
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 9 | -9.0 (27.9) | 1.0 (20.6) | 4.7 (20.7) | -1.7 (22.3)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 12: number analyzed (Participants) | 28 | 33 | 17 | 18
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 12 | -10.7 (23.5) | -7.4 (22.0) | -7.2 (21.1) | 4.3 (19.9)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 15: number analyzed (Participants) | 29 | 28 | 13 | 17
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 15 | -3.8 (27.7) | -0.6 (22.0) | -12.8 (14.9) | 4.6 (24.9)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 18: number analyzed (Participants) | 27 | 24 | 11 | 14
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 18 | -7.0 (24.1) | -8.3 (19.2) | -4.0 (13.4) | 5.6 (19.4)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 21: number analyzed (Participants) | 22 | 24 | 12 | 12
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 21 | -3.5 (20.7) | 3.0 (18.9) | -5.1 (18.0) | 6.5 (30.9)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 24: number analyzed (Participants) | 19 | 17 | 13 | 8
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 24 | -10.5 (20.1) | 0.7 (17.3) | -7.7 (16.0) | 4.2 (22.2)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 15 | 6 | 4
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 27 | -6.3 (24.2) | -1.9 (17.3) | -9.3 (14.8) | 22.2 (24.0)
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Speech Problems; Change from Baseline at Week 90 | -22.2 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Baseline: number analyzed (Participants) | 50 | 48 | 28 | 36
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Baseline | 33.8 (32.8) | 34.2 (28.5) | 28.3 (26.7) | 24.8 (26.7)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 3: number analyzed (Participants) | 40 | 38 | 22 | 28
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 3 | 0.7 (31.5) | 0.2 (24.8) | 7.4 (20.0) | 3.9 (14.1)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 6: number analyzed (Participants) | 29 | 34 | 16 | 26
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 6 | -9.2 (18.0) | -6.9 (33.0) | 3.0 (16.8) | 2.4 (25.8)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 9: number analyzed (Participants) | 25 | 27 | 19 | 21
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 9 | -8.2 (23.9) | 1.2 (24.4) | 4.4 (28.8) | -3.6 (17.4)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 12: number analyzed (Participants) | 29 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 12 | -4.9 (27.5) | -9.4 (24.2) | 2.5 (24.2) | 6.1 (15.4)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 15 | -3.0 (23.3) | -1.4 (32.9) | -3.4 (22.5) | 8.3 (20.0)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 18 | -9.2 (21.4) | 0.0 (30.8) | 3.5 (25.2) | 6.1 (24.7)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 23 | 12 | 13
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 21 | -8.0 (27.7) | 7.6 (28.7) | 4.6 (23.8) | -3.8 (20.0)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 16 | 13 | 9
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 24 | -17.1 (24.0) | -1.0 (20.4) | 1.7 (26.7) | 9.9 (23.3)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 14 | 6 | 5
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 27 | -3.6 (24.8) | -1.2 (13.8) | 0.5 (16.3) | 20.0 (19.2)
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Trouble with Social Eating; Change from Baseline at Week 90 | -8.3 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Baseline: number analyzed (Participants) | 51 | 49 | 28 | 37
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Baseline | 21.4 (24.6) | 21.7 (28.0) | 15.5 (22.2) | 13.4 (19.6)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 3: number analyzed (Participants) | 40 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 3 | -3.5 (24.4) | 5.4 (21.6) | 5.2 (19.9) | 6.9 (15.0)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 6: number analyzed (Participants) | 31 | 35 | 16 | 26
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 6 | -9.2 (13.9) | -2.7 (28.1) | 2.9 (22.4) | 10.0 (21.5)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 9 | -8.0 (17.6) | 1.4 (18.5) | 6.8 (24.8) | -0.6 (11.7)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 12: number analyzed (Participants) | 29 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 12 | -1.7 (18.0) | -5.4 (22.4) | -2.8 (19.0) | 2.5 (20.4)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 15 | 1.4 (28.6) | -2.1 (24.0) | -5.1 (15.7) | 7.0 (19.1)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 18 | -1.8 (24.6) | -1.6 (22.2) | -2.4 (18.7) | 0.4 (15.0)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 12 | 13
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 21 | -1.9 (26.9) | 9.3 (18.0) | -2.2 (20.4) | 9.2 (23.0)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 24 | -5.1 (22.3) | 2.7 (11.6) | 0.5 (23.2) | 5.2 (9.9)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 27 | -4.3 (25.8) | -0.9 (19.5) | -4.4 (15.6) | 17.3 (28.5)
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Trouble with Social Contact; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Less Sexuality; Baseline: number analyzed (Participants) | 51 | 45 | 27 | 34
  Parameter: Symptom Scales / Items: Less Sexuality; Baseline | 34.0 (34.8) | 38.9 (41.0) | 30.9 (29.1) | 40.2 (37.9)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 3: number analyzed (Participants) | 39 | 36 | 21 | 26
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 3 | 4.3 (23.5) | 7.4 (37.9) | 9.5 (38.6) | 4.5 (23.8)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 6: number analyzed (Participants) | 28 | 29 | 14 | 23
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 6 | 4.2 (28.9) | 16.1 (43.3) | 3.6 (39.9) | -3.6 (32.6)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 9: number analyzed (Participants) | 26 | 26 | 16 | 19
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 9 | 7.1 (42.2) | 5.1 (39.4) | 18.7 (43.4) | 1.8 (31.4)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 12: number analyzed (Participants) | 27 | 28 | 15 | 17
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 12 | 0.6 (32.2) | 5.4 (36.3) | 22.2 (40.7) | 2.9 (30.2)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 15: number analyzed (Participants) | 28 | 24 | 12 | 16
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 15 | 9.5 (43.4) | 9.0 (42.3) | 2.8 (48.6) | 2.1 (30.4)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 18: number analyzed (Participants) | 26 | 20 | 9 | 12
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 18 | -3.2 (33.7) | 2.5 (39.5) | 5.6 (39.1) | -5.6 (32.0)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 20 | 10 | 11
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 21 | -2.9 (42.8) | 0.8 (39.2) | 21.7 (36.9) | 3.0 (38.6)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 24: number analyzed (Participants) | 19 | 13 | 10 | 7
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 24 | -0.9 (23.9) | 7.7 (47.4) | 11.7 (27.3) | -9.5 (41.8)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 27: number analyzed (Participants) | 13 | 12 | 4 | 3
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 27 | 9.0 (23.2) | 6.9 (47.9) | -25.0 (50.0) | -33.3 (57.7)
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Less Sexuality; Change from Baseline at Week 90 | -33.3 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Teeth; Baseline: number analyzed (Participants) | 50 | 46 | 28 | 36
  Parameter: Symptom Scales / Items: Teeth; Baseline | 21.3 (33.5) | 16.7 (28.8) | 14.3 (32.0) | 30.6 (37.7)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 38 | 23 | 29
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 3 | -11.4 (36.2) | -0.9 (26.3) | 7.2 (24.5) | -11.5 (27.1)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 6: number analyzed (Participants) | 29 | 32 | 16 | 27
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 6 | -5.7 (25.3) | -8.3 (36.9) | 2.1 (14.8) | -17.3 (33.8)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 9: number analyzed (Participants) | 28 | 27 | 19 | 21
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 9 | 6.0 (28.8) | -2.5 (22.5) | -1.8 (36.0) | -17.5 (34.3)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 12: number analyzed (Participants) | 30 | 29 | 17 | 19
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 12 | 6.7 (34.4) | 1.1 (33.9) | 5.9 (29.4) | -8.8 (38.2)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 25 | 13 | 18
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 15 | 0.0 (31.6) | 5.3 (39.3) | -12.8 (29.0) | -9.3 (35.8)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 18: number analyzed (Participants) | 27 | 24 | 11 | 14
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 18 | 0.0 (29.2) | -1.4 (45.6) | 0.0 (14.9) | -16.7 (36.4)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 21: number analyzed (Participants) | 24 | 20 | 11 | 13
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 21 | 4.2 (30.0) | 10.0 (42.0) | 6.1 (13.5) | -5.1 (26.7)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 14 | 13 | 9
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 24 | 3.3 (37.3) | 4.8 (43.1) | 7.7 (20.0) | -22.2 (44.1)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 11 | 6 | 5
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 27 | 2.4 (24.3) | -6.1 (13.5) | 0.0 (21.1) | -20.0 (50.6)
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Teeth; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Opening Mouth; Baseline: number analyzed (Participants) | 50 | 48 | 28 | 37
  Parameter: Symptom Scales / Items: Opening Mouth; Baseline | 32.7 (40.7) | 39.6 (41.1) | 22.6 (32.8) | 37.8 (41.7)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 3 | -2.4 (34.5) | 3.3 (30.6) | 11.6 (21.6) | -4.6 (19.4)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 6: number analyzed (Participants) | 31 | 34 | 16 | 27
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 6 | -6.5 (33.8) | -11.8 (24.5) | 10.4 (26.4) | -6.2 (29.3)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 27 | 19 | 21
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 9 | 2.5 (34.5) | -6.2 (32.1) | 8.8 (36.6) | -4.8 (24.2)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 12: number analyzed (Participants) | 30 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 12 | -3.3 (35.4) | -9.4 (39.0) | 11.8 (23.4) | 0.0 (24.8)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 15: number analyzed (Participants) | 31 | 27 | 13 | 18
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 15 | 0.0 (38.5) | -8.6 (45.8) | 7.7 (14.6) | 1.9 (35.2)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 14
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 18 | 3.6 (26.2) | -6.7 (36.0) | 12.1 (16.8) | 2.4 (27.6)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 23 | 11 | 13
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 21 | 2.9 (26.4) | 1.4 (38.2) | 3.0 (10.1) | 0.0 (27.2)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 16 | 13 | 9
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 24 | 10.0 (28.8) | -2.1 (39.4) | 10.3 (21.0) | -3.7 (20.0)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 27 | 8.9 (23.5) | -16.7 (31.4) | 5.6 (13.6) | 20.0 (29.8)
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Opening Mouth; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Dry Mouth; Baseline | 42.3 (35.6) | 38.1 (36.0) | 34.5 (33.3) | 49.5 (37.4)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 3: number analyzed (Participants) | 42 | 42 | 23 | 29
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 3 | -9.5 (36.3) | -0.8 (26.0) | 0.0 (24.6) | -12.6 (32.6)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 6 | -9.4 (30.8) | 0.9 (34.3) | 2.1 (33.3) | -13.6 (29.6)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 9: number analyzed (Participants) | 28 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 9 | -7.1 (43.8) | -2.3 (28.1) | 1.8 (32.3) | -9.5 (39.6)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 12: number analyzed (Participants) | 32 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 12 | -3.1 (37.3) | -5.1 (40.9) | -3.9 (33.1) | -7.0 (17.8)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 15: number analyzed (Participants) | 31 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 15 | -5.4 (40.5) | -1.2 (41.1) | 2.6 (37.2) | -1.9 (31.3)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 18 | -8.3 (35.3) | -2.6 (38.8) | 6.1 (46.7) | -11.9 (21.1)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 21 | -4.2 (37.2) | 1.4 (44.5) | -3.0 (48.2) | -15.4 (29.2)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 24 | -4.8 (38.4) | -11.8 (37.2) | -10.3 (37.0) | -14.8 (29.4)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 27 | 0.0 (42.2) | -20.0 (32.9) | 0.0 (51.6) | 6.7 (36.5)
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Dry Mouth; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Sticky Saliva; Baseline: number analyzed (Participants) | 52 | 49 | 28 | 36
  Parameter: Symptom Scales / Items: Sticky Saliva; Baseline | 41.0 (35.9) | 44.9 (36.4) | 38.1 (36.0) | 45.4 (41.5)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 3: number analyzed (Participants) | 42 | 42 | 23 | 28
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 3 | -7.1 (35.7) | -5.6 (36.0) | 1.4 (40.8) | -1.2 (27.9)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 6 | -7.3 (23.5) | -8.3 (38.5) | 0.0 (29.8) | -1.2 (25.3)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 9 | -1.2 (38.7) | -10.3 (29.7) | -10.5 (35.2) | 3.2 (36.4)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 12: number analyzed (Participants) | 32 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 12 | -1.0 (35.4) | -10.1 (30.6) | -15.7 (41.0) | 7.0 (23.8)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 15: number analyzed (Participants) | 32 | 28 | 12 | 18
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 15 | -1.0 (26.1) | -11.9 (39.8) | -11.1 (35.8) | 0.0 (30.2)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 18 | -3.6 (33.1) | -10.3 (33.7) | -12.1 (45.4) | 2.4 (27.6)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 21 | 1.4 (31.8) | -12.5 (40.3) | -6.1 (41.7) | 5.1 (42.7)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 24 | -3.2 (29.6) | -13.7 (33.5) | -7.7 (45.4) | 3.7 (20.0)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 27 | 0.0 (24.3) | -26.7 (22.5) | -5.6 (49.1) | 20.0 (29.8)
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Sticky Saliva; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Coughing: Baseline | 31.4 (28.3) | 32.7 (35.7) | 41.7 (33.5) | 36.9 (30.2)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 3 | 0.0 (27.5) | 0.0 (26.9) | 2.9 (22.3) | 0.0 (34.5)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 6 | 0.0 (25.4) | -4.6 (40.0) | -6.3 (21.8) | 1.2 (31.3)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 9: number analyzed (Participants) | 28 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 9 | 3.6 (35.5) | 0.0 (33.3) | -1.8 (28.3) | -1.6 (24.7)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 12: number analyzed (Participants) | 32 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 12 | -5.2 (26.9) | -1.0 (38.6) | -7.8 (36.4) | 8.8 (31.1)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 15 | 4.3 (30.7) | -3.6 (38.9) | -2.6 (34.6) | -9.3 (25.1)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 26 | 11 | 14
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 18 | -4.8 (31.1) | 2.6 (37.6) | 0.0 (21.1) | 7.1 (26.7)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 21 | -1.4 (20.8) | 4.2 (31.6) | -6.1 (25.0) | 2.6 (34.6)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 24 | -1.6 (28.8) | 0.0 (16.7) | -17.9 (29.2) | 3.7 (26.1)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 27 | -2.1 (25.7) | -6.7 (36.1) | 0.0 (21.1) | 13.3 (38.0)
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Coughing: Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Felt Ill: Baseline: number analyzed (Participants) | 52 | 47 | 28 | 37
  Parameter: Symptom Scales / Items: Felt Ill: Baseline | 24.4 (31.0) | 31.9 (35.4) | 27.4 (27.3) | 22.5 (28.4)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 3: number analyzed (Participants) | 42 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 3 | 1.6 (30.3) | -2.4 (28.3) | 11.6 (25.8) | 5.7 (28.3)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 6: number analyzed (Participants) | 32 | 36 | 16 | 27
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 6 | -8.3 (29.3) | -13.0 (36.8) | 2.1 (19.1) | -1.2 (29.9)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 9: number analyzed (Participants) | 27 | 28 | 18 | 21
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 9 | 4.9 (30.2) | -10.7 (39.6) | -3.7 (22.5) | 0.0 (23.6)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 12: number analyzed (Participants) | 32 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 12 | 1.0 (28.7) | -9.4 (31.9) | -2.0 (30.0) | -1.8 (28.3)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 15: number analyzed (Participants) | 31 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 15 | 5.4 (31.1) | -15.5 (36.8) | 2.6 (28.7) | 5.6 (34.8)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 14
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 18 | 3.6 (24.6) | -10.7 (36.9) | 9.1 (15.6) | 0.0 (29.2)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 13
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 21 | 4.2 (17.9) | 5.6 (32.1) | 12.1 (27.0) | 10.3 (41.7)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 24: number analyzed (Participants) | 21 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 24 | 3.2 (20.8) | -2.0 (27.6) | 7.7 (20.0) | 11.1 (37.3)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 27: number analyzed (Participants) | 16 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 27 | 10.4 (31.5) | -4.4 (27.8) | 5.6 (13.6) | -13.3 (38.0)
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Felt Ill: Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Pain Killers; Baseline: number analyzed (Participants) | 51 | 49 | 28 | 37
  Parameter: Symptom Scales / Items: Pain Killers; Baseline | 78.4 (41.5) | 75.5 (43.4) | 78.6 (41.8) | 78.4 (41.7)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 42 | 23 | 28
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 3 | 7.3 (34.6) | 7.1 (46.3) | 0.0 (52.2) | 3.6 (42.9)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 6: number analyzed (Participants) | 31 | 36 | 16 | 26
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 6 | -12.9 (42.8) | -8.3 (55.4) | 6.3 (68.0) | -11.5 (58.8)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 9 | -14.8 (45.6) | 3.4 (32.5) | -10.5 (56.7) | -14.3 (47.8)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 12: number analyzed (Participants) | 30 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 12 | -20.0 (48.4) | -9.1 (52.2) | -17.6 (52.9) | 0.0 (33.3)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 15 | -16.7 (64.8) | -7.1 (46.6) | -30.8 (75.1) | -11.1 (47.1)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 18 | -21.4 (63.0) | -4.0 (45.5) | 0.0 (77.5) | -13.3 (51.6)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 12 | 13
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 21 | -30.4 (63.5) | -12.5 (53.7) | -33.3 (65.1) | -15.4 (37.6)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 16 | 13 | 9
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 24 | -30.0 (57.1) | -25.0 (44.7) | -23.1 (59.9) | -22.2 (44.1)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 27 | -35.7 (63.3) | -13.3 (51.6) | -33.3 (51.6) | -20.0 (44.7)
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Pain Killers; Change from Baseline at Week 90 | -100.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Nutritional Supplements; Baseline: number analyzed (Participants) | 50 | 48 | 28 | 37
  Parameter: Symptom Scales / Items: Nutritional Supplements; Baseline | 34.0 (47.9) | 47.9 (50.5) | 42.9 (50.4) | 48.6 (50.7)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 3 | 4.9 (44.4) | 12.2 (51.0) | 13.0 (45.8) | 0.0 (53.5)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 6: number analyzed (Participants) | 31 | 36 | 16 | 25
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 6 | -9.7 (53.9) | -5.6 (58.3) | 6.3 (57.4) | -12.0 (52.6)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 28 | 19 | 20
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 9 | 3.7 (64.9) | -7.1 (66.3) | 0.0 (57.7) | 5.0 (60.5)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 12: number analyzed (Participants) | 29 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 12 | 17.2 (65.8) | -6.3 (56.4) | 0.0 (50.0) | -15.8 (50.1)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 27 | 13 | 18
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 15 | 3.3 (61.5) | -3.7 (58.7) | -15.4 (55.5) | -11.1 (47.1)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 24 | 11 | 15
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 18 | -7.1 (60.4) | -4.2 (62.4) | 0.0 (44.7) | 6.7 (59.4)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 23 | 12 | 13
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 21 | 4.3 (63.8) | 4.3 (63.8) | 16.7 (57.7) | 23.1 (59.9)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 24 | 15.0 (48.9) | 11.8 (69.7) | -15.4 (55.5) | -11.1 (60.1)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 14 | 6 | 5
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 27 | 14.3 (36.3) | 7.1 (82.9) | -16.7 (40.8) | 0.0 (70.7)
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Nutritional Supplements; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Feeding Tube; Baseline: number analyzed (Participants) | 50 | 48 | 28 | 37
  Parameter: Symptom Scales / Items: Feeding Tube; Baseline | 28.0 (45.4) | 27.1 (44.9) | 28.6 (46.0) | 32.4 (47.5)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 3: number analyzed (Participants) | 41 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 3 | 4.9 (38.4) | 4.9 (21.8) | 4.3 (20.9) | -6.9 (25.8)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 6: number analyzed (Participants) | 31 | 35 | 15 | 26
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 6 | 0.0 (25.8) | -5.7 (33.8) | -6.7 (25.8) | -7.7 (39.2)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 28 | 19 | 21
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 9 | -11.1 (32.0) | 7.1 (26.2) | 5.3 (40.5) | -4.8 (38.4)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 12: number analyzed (Participants) | 29 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 12 | -3.4 (32.5) | 6.1 (34.8) | -5.9 (42.9) | 0.0 (33.3)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 27 | 13 | 18
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 15 | 3.3 (32.0) | 0.0 (27.7) | -7.7 (49.4) | 5.6 (23.6)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 23 | 11 | 15
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 18 | -3.6 (33.1) | 4.3 (20.9) | -9.1 (30.2) | 0.0 (37.8)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 23 | 12 | 13
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 21 | -4.3 (36.7) | 4.3 (20.9) | -16.7 (38.9) | 7.7 (27.7)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 24 | 0.0 (32.4) | 5.9 (24.3) | -15.4 (37.6) | 0.0 (0.0)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 13 | 6 | 5
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 27 | 0.0 (0.0) | 7.7 (27.7) | -16.7 (40.8) | 0.0 (0.0)
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Feeding Tube; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Weight Loss; Baseline: number analyzed (Participants) | 50 | 49 | 28 | 37
  Parameter: Symptom Scales / Items: Weight Loss; Baseline | 32.0 (47.1) | 44.9 (50.3) | 28.6 (46.0) | 29.7 (46.3)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 3: number analyzed (Participants) | 39 | 41 | 23 | 29
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 3 | 23.1 (62.7) | -4.9 (59.0) | 30.4 (55.9) | 10.3 (61.8)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 6: number analyzed (Participants) | 30 | 36 | 16 | 26
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 6 | -6.7 (74.0) | -13.9 (59.3) | 12.5 (50.0) | 19.2 (63.4)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 9: number analyzed (Participants) | 27 | 29 | 19 | 21
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 9 | 3.7 (70.6) | -17.2 (60.2) | 0.0 (57.7) | -9.5 (53.9)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 12: number analyzed (Participants) | 29 | 33 | 17 | 19
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 12 | -17.2 (46.8) | -18.2 (58.4) | 11.8 (33.2) | -5.3 (52.4)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 17
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 15 | 13.3 (73.0) | -10.7 (73.7) | 15.4 (37.6) | -5.9 (65.9)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 18: number analyzed (Participants) | 28 | 25 | 11 | 15
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 18 | 0.0 (60.9) | -20.0 (57.7) | 0.0 (44.7) | 6.7 (59.4)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 21: number analyzed (Participants) | 23 | 24 | 12 | 13
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 21 | 4.3 (47.5) | -4.2 (75.1) | 25.0 (45.2) | 7.7 (76.0)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 24: number analyzed (Participants) | 20 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 24 | -5.0 (39.4) | -5.9 (65.9) | 7.7 (49.4) | 33.3 (50.0)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 27 | 0.0 (55.5) | -13.3 (74.3) | 0.0 (0.0) | 40.0 (54.8)
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Weight Loss; Change from Baseline at Week 90 | 0.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |
  Parameter: Symptom Scales / Items: Weight Gain; Baseline: number analyzed (Participants) | 49 | 49 | 28 | 37
  Parameter: Symptom Scales / Items: Weight Gain; Baseline | 14.3 (35.4) | 8.2 (27.7) | 21.4 (41.8) | 18.9 (39.7)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 3: number analyzed (Participants) | 39 | 40 | 23 | 29
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 3 | 7.7 (53.2) | 27.5 (55.4) | 4.3 (36.7) | -6.9 (53.0)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 6: number analyzed (Participants) | 30 | 36 | 16 | 26
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 6 | 10.0 (54.8) | 25.0 (43.9) | 0.0 (63.2) | 7.7 (48.4)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 9: number analyzed (Participants) | 26 | 28 | 18 | 21
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 9 | 3.8 (59.9) | 14.3 (44.8) | 5.6 (63.9) | 19.0 (60.2)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 12: number analyzed (Participants) | 28 | 32 | 17 | 19
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 12 | 14.3 (52.5) | 6.3 (50.4) | 23.5 (43.7) | 26.3 (56.2)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 15: number analyzed (Participants) | 30 | 28 | 13 | 18
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 15 | 6.7 (58.3) | 25.0 (64.5) | 0.0 (40.8) | 11.1 (47.1)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 18: number analyzed (Participants) | 27 | 24 | 11 | 15
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 18 | 7.4 (38.5) | 16.7 (56.5) | -18.2 (60.3) | 6.7 (59.4)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 21: number analyzed (Participants) | 22 | 24 | 12 | 13
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 21 | 18.2 (39.5) | 4.2 (55.0) | 0.0 (73.9) | 15.4 (68.9)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 24: number analyzed (Participants) | 19 | 17 | 13 | 9
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 24 | 21.1 (63.1) | 17.6 (52.9) | 0.0 (40.8) | 11.1 (60.1)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 27: number analyzed (Participants) | 14 | 15 | 6 | 5
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 27 | 28.6 (61.1) | 33.3 (61.7) | -16.7 (40.8) | 20.0 (44.7)
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Parameter: Symptom Scales / Items: Weight Gain; Change from Baseline at Week 90 | -100.0 (NA) — The Standard Deviation can not be calculated for one participant. |  |  |

14. Secondary Outcome: Phase 2 Cohorts: Number of Participants With 5-level EuroQol 5 Dimensions Questionnaire (EQ-5D-5L) Score
Description: EQ-5D-5L was an instrument for use as a measure of health outcome. The EQ-5D-5L consisted of 2 sections: EuroQoL (5 dimensions) (EQ-5D) descriptive system and the EuroQoL visual analogue scale (EQ-VAS). EQ-5D comprised the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Number of participants per category are reported.
Time Frame: Baseline, Week 3, Week 6, Week 9, Week 12, Week 15, Week 18, Week 21, Week 24, Week 27 and Week 90
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum+5-FU: Participants received magrolimab + zimberelimab + platinum + 5 FU IV infusions as mentioned below:
  Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, beginning at Day 8 and for the next 5 doses (Cycle 1 Days 8, 15, and Cycle 2 Days 1, 8 and 15); 60 mg/kg, starting Cycle 3 Day 1 onwards for every 21-day cycle for up to 37 weeks; Zimberelimab 360 mg IV on Day 1 of every 21-day cycle for up to 40 weeks; 5-FU 1000 mg/m^2/day continuous IV On Day 1 to 4 of Cycles 1 to 6 for 21-day cycle each for up to 19 weeks; Cisplatin 100 mg/m^2 IV or Carboplatin AUC 5 IV on Day 1 of Cycles 1 to 6 for 21-day cycle each for up to 18 weeks for carboplatin and 16 weeks for cisplatin.
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum+5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum+5-FU | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 51 | 50 | 27 | 36
Participants
  Mobility: Baseline: No Problems | 35 | 31 | 19 | 18
  Mobility: Baseline: Slight Problems | 9 | 10 | 4 | 7
  Mobility: Baseline: Moderate Problems | 5 | 7 | 2 | 9
  Mobility: Baseline: Severe Problems | 2 | 1 | 2 | 2
  Mobility: Baseline: Extreme Problems | 0 | 1 | 0 | 0
  Mobility: Week 3: number analyzed (Participants) | 42 | 43 | 23 | 30
  Mobility: Week 3: No Problems | 29 | 28 | 13 | 16
  Mobility: Week 3: Slight Problems | 7 | 10 | 5 | 6
  Mobility: Week 3: Moderate Problems | 4 | 3 | 3 | 5
  Mobility: Week 3: Severe Problems | 2 | 2 | 2 | 2
  Mobility: Week 3: Extreme Problems | 0 | 0 | 0 | 1
  Mobility: Week 6: number analyzed (Participants) | 30 | 40 | 16 | 27
  Mobility: Week 6: No Problems | 17 | 28 | 11 | 12
  Mobility: Week 6: Slight Problems | 7 | 9 | 3 | 8
  Mobility: Week 6: Moderate Problems | 3 | 1 | 2 | 4
  Mobility: Week 6: Severe Problems | 1 | 1 | 0 | 2
  Mobility: Week 6: Extreme Problems | 2 | 1 | 0 | 1
  Mobility: Week 9: number analyzed (Participants) | 29 | 30 | 19 | 21
  Mobility: Week 9: No Problems | 19 | 21 | 12 | 12
  Mobility: Week 9: Slight Problems | 5 | 5 | 5 | 4
  Mobility: Week 9: Moderate Problems | 4 | 2 | 1 | 4
  Mobility: Week 9: Severe Problems | 1 | 1 | 1 | 1
  Mobility: Week 9: Extreme Problems | 0 | 1 | 0 | 0
  Mobility: Week 12: number analyzed (Participants) | 31 | 34 | 18 | 19
  Mobility: Week 12: No Problems | 18 | 22 | 12 | 11
  Mobility: Week 12: Slight Problems | 9 | 6 | 4 | 4
  Mobility: Week 12: Moderate Problems | 2 | 4 | 2 | 3
  Mobility: Week 12: Severe Problems | 1 | 1 | 0 | 0
  Mobility: Week 12: Extreme Problems | 1 | 1 | 0 | 1
  Mobility: Week 15: number analyzed (Participants) | 31 | 31 | 12 | 18
  Mobility: Week 15: No Problems | 22 | 17 | 9 | 9
  Mobility: Week 15: Slight Problems | 5 | 7 | 2 | 5
  Mobility: Week 15: Moderate Problems | 1 | 5 | 0 | 2
  Mobility: Week 15: Severe Problems | 3 | 1 | 1 | 2
  Mobility: Week 15: Extreme Problems | 0 | 1 | 0 | 0
  Mobility: Week 18: number analyzed (Participants) | 29 | 24 | 11 | 16
  Mobility: Week 18: No Problems | 19 | 18 | 10 | 5
  Mobility: Week 18: Slight Problems | 5 | 3 | 1 | 7
  Mobility: Week 18: Moderate Problems | 2 | 1 | 0 | 2
  Mobility: Week 18: Severe Problems | 3 | 2 | 0 | 2
  Mobility: Week 18: Extreme Problems | 0 | 0 | 0 | 0
  Mobility: Week 21: number analyzed (Participants) | 24 | 24 | 13 | 12
  Mobility: Week 21: No Problems | 15 | 11 | 9 | 2
  Mobility: Week 21: Slight Problems | 6 | 8 | 1 | 6
  Mobility: Week 21: Moderate Problems | 2 | 3 | 1 | 3
  Mobility: Week 21: Severe Problems | 1 | 0 | 1 | 1
  Mobility: Week 21: Extreme Problems | 0 | 2 | 1 | 0
  Mobility: Week 24: number analyzed (Participants) | 21 | 18 | 13 | 8
  Mobility: Week 24: No Problems | 15 | 5 | 11 | 3
  Mobility: Week 24: Slight Problems | 4 | 8 | 0 | 0
  Mobility: Week 24: Moderate Problems | 1 | 4 | 2 | 4
  Mobility: Week 24: Severe Problems | 1 | 1 | 0 | 1
  Mobility: Week 24: Extreme Problems | 0 | 0 | 0 | 0
  Mobility: Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Mobility: Week 27: No Problems | 9 | 7 | 5 | 1
  Mobility: Week 27: Slight Problems | 4 | 5 | 1 | 0
  Mobility: Week 27: Moderate Problems | 2 | 0 | 0 | 3
  Mobility: Week 27: Severe Problems | 0 | 2 | 0 | 1
  Mobility: Week 27: Extreme Problems | 0 | 0 | 0 | 0
  Mobility: Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Mobility: Week 90: No Problems | 1 |  |  |
  Mobility: Week 90: Slight Problems | 0 |  |  |
  Mobility: Week 90: Moderate Problems | 0 |  |  |
  Mobility: Week 90: Severe Problems | 0 |  |  |
  Mobility: Week 90: Extreme Problems | 0 |  |  |
  Self-Care: Baseline: number analyzed (Participants) | 50 | 49 | 27 | 36
  Self-Care: Baseline: No Problems | 38 | 38 | 23 | 30
  Self-Care: Baseline: Slight Problems | 6 | 8 | 3 | 3
  Self-Care: Baseline: Moderate Problems | 3 | 2 | 0 | 2
  Self-Care: Baseline: Severe Problems | 3 | 0 | 1 | 1
  Self-Care: Baseline: Extreme Problems | 0 | 1 | 0 | 0
  Self-Care: Week 3: number analyzed (Participants) | 42 | 43 | 23 | 30
  Self-Care: Week 3: No Problems | 31 | 32 | 16 | 21
  Self-Care: Week 3: Slight Problems | 5 | 7 | 5 | 5
  Self-Care: Week 3: Moderate Problems | 5 | 4 | 0 | 2
  Self-Care: Week 3: Severe Problems | 1 | 0 | 2 | 2
  Self-Care: Week 3: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 6: number analyzed (Participants) | 30 | 40 | 16 | 27
  Self-Care: Week 6: No Problems | 25 | 34 | 13 | 19
  Self-Care: Week 6: Slight Problems | 3 | 3 | 3 | 6
  Self-Care: Week 6: Moderate Problems | 1 | 1 | 0 | 0
  Self-Care: Week 6: Severe Problems | 0 | 2 | 0 | 2
  Self-Care: Week 6: Extreme Problems | 1 | 0 | 0 | 0
  Self-Care: Week 9: number analyzed (Participants) | 29 | 30 | 19 | 21
  Self-Care: Week 9: No Problems | 22 | 24 | 16 | 17
  Self-Care: Week 9: Slight Problems | 5 | 4 | 2 | 3
  Self-Care: Week 9: Moderate Problems | 2 | 1 | 0 | 1
  Self-Care: Week 9: Severe Problems | 0 | 1 | 1 | 0
  Self-Care: Week 9: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 12: number analyzed (Participants) | 31 | 34 | 18 | 19
  Self-Care: Week 12: No Problems | 24 | 27 | 15 | 17
  Self-Care: Week 12: Slight Problems | 5 | 3 | 2 | 1
  Self-Care: Week 12: Moderate Problems | 0 | 4 | 1 | 0
  Self-Care: Week 12: Severe Problems | 2 | 0 | 0 | 1
  Self-Care: Week 12: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 15: number analyzed (Participants) | 31 | 31 | 12 | 18
  Self-Care: Week 15: No Problems | 24 | 25 | 10 | 13
  Self-Care: Week 15: Slight Problems | 4 | 4 | 1 | 5
  Self-Care: Week 15: Moderate Problems | 2 | 1 | 1 | 0
  Self-Care: Week 15: Severe Problems | 1 | 1 | 0 | 0
  Self-Care: Week 15: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 18: number analyzed (Participants) | 29 | 24 | 11 | 16
  Self-Care: Week 18: No Problems | 22 | 21 | 10 | 13
  Self-Care: Week 18: Slight Problems | 4 | 2 | 1 | 2
  Self-Care: Week 18: Moderate Problems | 1 | 0 | 0 | 1
  Self-Care: Week 18: Severe Problems | 2 | 1 | 0 | 0
  Self-Care: Week 18: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 21: number analyzed (Participants) | 24 | 24 | 13 | 12
  Self-Care: Week 21: No Problems | 18 | 17 | 12 | 8
  Self-Care: Week 21: Slight Problems | 4 | 5 | 1 | 2
  Self-Care: Week 21: Moderate Problems | 1 | 1 | 0 | 2
  Self-Care: Week 21: Severe Problems | 0 | 0 | 0 | 0
  Self-Care: Week 21: Extreme Problems | 1 | 1 | 0 | 0
  Self-Care: Week 24: number analyzed (Participants) | 21 | 18 | 13 | 8
  Self-Care: Week 24: No Problems | 17 | 15 | 11 | 6
  Self-Care: Week 24: Slight Problems | 2 | 0 | 1 | 0
  Self-Care: Week 24: Moderate Problems | 2 | 2 | 1 | 2
  Self-Care: Week 24: Severe Problems | 0 | 1 | 0 | 0
  Self-Care: Week 24: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Self-Care: Week 27: No Problems | 12 | 12 | 6 | 3
  Self-Care: Week 27: Slight Problems | 1 | 1 | 0 | 1
  Self-Care: Week 27: Moderate Problems | 2 | 0 | 0 | 1
  Self-Care: Week 27: Severe Problems | 0 | 1 | 0 | 0
  Self-Care: Week 27: Extreme Problems | 0 | 0 | 0 | 0
  Self-Care: Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Self-Care: Week 90: No Problems | 1 |  |  |
  Self-Care: Week 90: Slight Problems | 0 |  |  |
  Self-Care: Week 90: Moderate Problems | 0 |  |  |
  Self-Care: Week 90: Severe Problems | 0 |  |  |
  Self-Care: Week 90: Extreme Problems | 0 |  |  |
  Usual Activities: Baseline: number analyzed (Participants) | 51 | 49 | 26 | 36
  Usual Activities: Baseline: No Problems | 25 | 24 | 14 | 15
  Usual Activities: Baseline: Slight Problems | 13 | 14 | 9 | 12
  Usual Activities: Baseline: Moderate Problems | 8 | 7 | 1 | 3
  Usual Activities: Baseline: Severe Problems | 4 | 1 | 2 | 2
  Usual Activities: Baseline: Extreme Problems | 1 | 3 | 0 | 4
  Usual Activities: Week 3: number analyzed (Participants) | 42 | 42 | 23 | 30
  Usual Activities: Week 3: No Problems | 16 | 19 | 8 | 10
  Usual Activities: Week 3: Slight Problems | 17 | 15 | 9 | 11
  Usual Activities: Week 3: Moderate Problems | 5 | 6 | 4 | 7
  Usual Activities: Week 3: Severe Problems | 3 | 2 | 1 | 1
  Usual Activities: Week 3: Extreme Problems | 1 | 0 | 1 | 1
  Usual Activities: Week 6: number analyzed (Participants) | 30 | 40 | 16 | 27
  Usual Activities: Week 6: No Problems | 16 | 21 | 8 | 12
  Usual Activities: Week 6: Slight Problems | 10 | 12 | 3 | 4
  Usual Activities: Week 6: Moderate Problems | 2 | 5 | 5 | 5
  Usual Activities: Week 6: Severe Problems | 1 | 1 | 0 | 4
  Usual Activities: Week 6: Extreme Problems | 1 | 1 | 0 | 2
  Usual Activities: Week 9: number analyzed (Participants) | 29 | 30 | 19 | 21
  Usual Activities: Week 9: No Problems | 14 | 19 | 10 | 11
  Usual Activities: Week 9: Slight Problems | 11 | 4 | 3 | 7
  Usual Activities: Week 9: Moderate Problems | 4 | 5 | 6 | 1
  Usual Activities: Week 9: Severe Problems | 0 | 2 | 0 | 2
  Usual Activities: Week 9: Extreme Problems | 0 | 0 | 0 | 0
  Usual Activities: Week 12: number analyzed (Participants) | 31 | 33 | 18 | 19
  Usual Activities: Week 12: No Problems | 16 | 21 | 13 | 9
  Usual Activities: Week 12: Slight Problems | 10 | 8 | 3 | 7
  Usual Activities: Week 12: Moderate Problems | 1 | 3 | 2 | 2
  Usual Activities: Week 12: Severe Problems | 2 | 0 | 0 | 1
  Usual Activities: Week 12: Extreme Problems | 2 | 1 | 0 | 0
  Usual Activities: Week 15: number analyzed (Participants) | 30 | 30 | 12 | 18
  Usual Activities: Week 15: No Problems | 15 | 15 | 6 | 7
  Usual Activities: Week 15: Slight Problems | 8 | 8 | 4 | 7
  Usual Activities: Week 15: Moderate Problems | 5 | 5 | 2 | 2
  Usual Activities: Week 15: Severe Problems | 2 | 1 | 0 | 0
  Usual Activities: Week 15: Extreme Problems | 0 | 1 | 0 | 2
  Usual Activities: Week 18: number analyzed (Participants) | 29 | 24 | 11 | 16
  Usual Activities: Week 18: No Problems | 18 | 15 | 7 | 5
  Usual Activities: Week 18: Slight Problems | 6 | 7 | 4 | 8
  Usual Activities: Week 18: Moderate Problems | 2 | 2 | 0 | 1
  Usual Activities: Week 18: Severe Problems | 2 | 0 | 0 | 2
  Usual Activities: Week 18: Extreme Problems | 1 | 0 | 0 | 0
  Usual Activities: Week 21: number analyzed (Participants) | 24 | 23 | 13 | 12
  Usual Activities: Week 21: No Problems | 15 | 11 | 8 | 2
  Usual Activities: Week 21: Slight Problems | 9 | 9 | 1 | 4
  Usual Activities: Week 21: Moderate Problems | 0 | 2 | 2 | 5
  Usual Activities: Week 21: Severe Problems | 0 | 0 | 1 | 0
  Usual Activities: Week 21: Extreme Problems | 0 | 1 | 1 | 1
  Usual Activities: Week 24: number analyzed (Participants) | 21 | 17 | 13 | 7
  Usual Activities: Week 24: No Problems | 12 | 10 | 7 | 2
  Usual Activities: Week 24: Slight Problems | 5 | 4 | 3 | 2
  Usual Activities: Week 24: Moderate Problems | 2 | 1 | 3 | 3
  Usual Activities: Week 24: Severe Problems | 1 | 2 | 0 | 0
  Usual Activities: Week 24: Extreme Problems | 1 | 0 | 0 | 0
  Usual Activities: Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Usual Activities: Week 27: No Problems | 8 | 8 | 4 | 1
  Usual Activities: Week 27: Slight Problems | 4 | 3 | 2 | 0
  Usual Activities: Week 27: Moderate Problems | 3 | 1 | 0 | 3
  Usual Activities: Week 27: Severe Problems | 0 | 2 | 0 | 1
  Usual Activities: Week 27: Extreme Problems | 0 | 0 | 0 | 0
  Usual Activities: Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Usual Activities: Week 90: No Problems | 1 |  |  |
  Usual Activities: Week 90: Slight Problems | 0 |  |  |
  Usual Activities: Week 90: Moderate Problems | 0 |  |  |
  Usual Activities: Week 90: Severe Problems | 0 |  |  |
  Usual Activities: Week 90: Extreme Problems | 0 |  |  |
  Pain/Discomfort: Baseline: No Problems | 9 | 10 | 4 | 7
  Pain/Discomfort: Baseline: Slight Problems | 19 | 16 | 8 | 12
  Pain/Discomfort: Baseline: Moderate Problems | 15 | 15 | 11 | 12
  Pain/Discomfort: Baseline: Severe Problems | 6 | 8 | 2 | 5
  Pain/Discomfort: Baseline: Extreme Problems | 2 | 1 | 2 | 0
  Pain/Discomfort: Week 3: number analyzed (Participants) | 42 | 43 | 23 | 30
  Pain/Discomfort: Week 3: No Problems | 12 | 12 | 5 | 7
  Pain/Discomfort: Week 3: Slight Problems | 17 | 12 | 5 | 9
  Pain/Discomfort: Week 3: Moderate Problems | 10 | 15 | 7 | 10
  Pain/Discomfort: Week 3: Severe Problems | 3 | 4 | 5 | 4
  Pain/Discomfort: Week 3: Extreme Problems | 0 | 0 | 1 | 0
  Pain/Discomfort: Week 6: number analyzed (Participants) | 30 | 40 | 16 | 27
  Pain/Discomfort: Week 6: No Problems | 10 | 16 | 4 | 6
  Pain/Discomfort: Week 6: Slight Problems | 15 | 10 | 7 | 10
  Pain/Discomfort: Week 6: Moderate Problems | 5 | 11 | 4 | 8
  Pain/Discomfort: Week 6: Severe Problems | 0 | 3 | 1 | 3
  Pain/Discomfort: Week 6: Extreme Problems | 0 | 0 | 0 | 0
  Pain/Discomfort: Week 9: number analyzed (Participants) | 29 | 30 | 19 | 21
  Pain/Discomfort: Week 9: No Problems | 10 | 10 | 6 | 7
  Pain/Discomfort: Week 9: Slight Problems | 9 | 9 | 7 | 5
  Pain/Discomfort: Week 9: Moderate Problems | 8 | 8 | 5 | 8
  Pain/Discomfort: Week 9: Severe Problems | 2 | 3 | 1 | 0
  Pain/Discomfort: Week 9: Extreme Problems | 0 | 0 | 0 | 1
  Pain/Discomfort: Week 12: number analyzed (Participants) | 31 | 34 | 18 | 19
  Pain/Discomfort: Week 12: No Problems | 11 | 11 | 10 | 6
  Pain/Discomfort: Week 12: Slight Problems | 11 | 15 | 4 | 4
  Pain/Discomfort: Week 12: Moderate Problems | 5 | 6 | 3 | 8
  Pain/Discomfort: Week 12: Severe Problems | 3 | 1 | 1 | 0
  Pain/Discomfort: Week 12: Extreme Problems | 1 | 1 | 0 | 1
  Pain/Discomfort: Week 15: number analyzed (Participants) | 31 | 31 | 12 | 18
  Pain/Discomfort: Week 15: No Problems | 10 | 11 | 4 | 4
  Pain/Discomfort: Week 15: Slight Problems | 13 | 7 | 5 | 6
  Pain/Discomfort: Week 15: Moderate Problems | 5 | 9 | 3 | 8
  Pain/Discomfort: Week 15: Severe Problems | 3 | 3 | 0 | 0
  Pain/Discomfort: Week 15: Extreme Problems | 0 | 1 | 0 | 0
  Pain/Discomfort: Week 18: number analyzed (Participants) | 29 | 24 | 11 | 16
  Pain/Discomfort: Week 18: No Problems | 10 | 11 | 4 | 5
  Pain/Discomfort: Week 18: Slight Problems | 11 | 8 | 3 | 7
  Pain/Discomfort: Week 18: Moderate Problems | 8 | 5 | 4 | 2
  Pain/Discomfort: Week 18: Severe Problems | 0 | 0 | 0 | 2
  Pain/Discomfort: Week 18: Extreme Problems | 0 | 0 | 0 | 0
  Pain/Discomfort: Week 21: number analyzed (Participants) | 24 | 24 | 13 | 12
  Pain/Discomfort: Week 21: No Problems | 9 | 11 | 8 | 3
  Pain/Discomfort: Week 21: Slight Problems | 7 | 4 | 2 | 3
  Pain/Discomfort: Week 21: Moderate Problems | 5 | 6 | 3 | 5
  Pain/Discomfort: Week 21: Severe Problems | 3 | 3 | 0 | 1
  Pain/Discomfort: Week 21: Extreme Problems | 0 | 0 | 0 | 0
  Pain/Discomfort: Week 24: number analyzed (Participants) | 21 | 18 | 13 | 8
  Pain/Discomfort: Week 24: No Problems | 7 | 7 | 5 | 3
  Pain/Discomfort: Week 24: Slight Problems | 7 | 4 | 6 | 1
  Pain/Discomfort: Week 24: Moderate Problems | 7 | 6 | 1 | 3
  Pain/Discomfort: Week 24: Severe Problems | 0 | 0 | 0 | 1
  Pain/Discomfort: Week 24: Extreme Problems | 0 | 1 | 1 | 0
  Pain/Discomfort: Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Pain/Discomfort: Week 27: No Problems | 9 | 9 | 4 | 1
  Pain/Discomfort: Week 27: Slight Problems | 1 | 0 | 2 | 1
  Pain/Discomfort: Week 27: Moderate Problems | 4 | 2 | 0 | 2
  Pain/Discomfort: Week 27: Severe Problems | 1 | 3 | 0 | 0
  Pain/Discomfort: Week 27: Extreme Problems | 0 | 0 | 0 | 1
  Pain/Discomfort: Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Pain/Discomfort: Week 90: No Problems | 0 |  |  |
  Pain/Discomfort: Week 90: Slight Problems | 1 |  |  |
  Pain/Discomfort: Week 90: Moderate Problems | 0 |  |  |
  Pain/Discomfort: Week 90: Severe Problems | 0 |  |  |
  Pain/Discomfort: Week 90: Extreme Problems | 0 |  |  |
  Anxiety/Depression: Baseline: No Problems | 20 | 21 | 9 | 22
  Anxiety/Depression: Baseline: Slight Problems | 20 | 15 | 12 | 9
  Anxiety/Depression: Baseline: Moderate Problems | 6 | 8 | 5 | 5
  Anxiety/Depression: Baseline: Severe Problems | 4 | 3 | 1 | 0
  Anxiety/Depression: Baseline: Extreme Problems | 1 | 3 | 0 | 0
  Anxiety/Depression: Week 3: number analyzed (Participants) | 42 | 43 | 23 | 30
  Anxiety/Depression: Week 3: No Problems | 21 | 23 | 8 | 16
  Anxiety/Depression: Week 3: Slight Problems | 15 | 7 | 11 | 10
  Anxiety/Depression: Week 3: Moderate Problems | 3 | 9 | 3 | 3
  Anxiety/Depression: Week 3: Severe Problems | 3 | 4 | 1 | 1
  Anxiety/Depression: Week 3: Extreme Problems | 0 | 0 | 0 | 0
  Anxiety/Depression: Week 6: number analyzed (Participants) | 30 | 40 | 16 | 27
  Anxiety/Depression: Week 6: No Problems | 16 | 19 | 8 | 13
  Anxiety/Depression: Week 6: Slight Problems | 13 | 10 | 5 | 8
  Anxiety/Depression: Week 6: Moderate Problems | 1 | 7 | 3 | 5
  Anxiety/Depression: Week 6: Severe Problems | 0 | 3 | 0 | 1
  Anxiety/Depression: Week 6: Extreme Problems | 0 | 1 | 0 | 0
  Anxiety/Depression: Week 9: number analyzed (Participants) | 29 | 30 | 19 | 21
  Anxiety/Depression: Week 9: No Problems | 8 | 18 | 8 | 11
  Anxiety/Depression: Week 9: Slight Problems | 15 | 8 | 9 | 8
  Anxiety/Depression: Week 9: Moderate Problems | 6 | 3 | 2 | 2
  Anxiety/Depression: Week 9: Severe Problems | 0 | 0 | 0 | 0
  Anxiety/Depression: Week 9: Extreme Problems | 0 | 1 | 0 | 0
  Anxiety/Depression: Week 12: number analyzed (Participants) | 31 | 34 | 18 | 19
  Anxiety/Depression: Week 12: No Problems | 14 | 15 | 9 | 9
  Anxiety/Depression: Week 12: Slight Problems | 14 | 15 | 9 | 9
  Anxiety/Depression: Week 12: Moderate Problems | 0 | 4 | 0 | 1
  Anxiety/Depression: Week 12: Severe Problems | 1 | 0 | 0 | 0
  Anxiety/Depression: Week 12: Extreme Problems | 2 | 0 | 0 | 0
  Anxiety/Depression: Week 15: number analyzed (Participants) | 31 | 31 | 12 | 18
  Anxiety/Depression: Week 15: No Problems | 15 | 14 | 6 | 10
  Anxiety/Depression: Week 15: Slight Problems | 11 | 6 | 5 | 4
  Anxiety/Depression: Week 15: Moderate Problems | 3 | 8 | 1 | 4
  Anxiety/Depression: Week 15: Severe Problems | 1 | 3 | 0 | 0
  Anxiety/Depression: Week 15: Extreme Problems | 1 | 0 | 0 | 0
  Anxiety/Depression: Week 18: number analyzed (Participants) | 29 | 24 | 10 | 15
  Anxiety/Depression: Week 18: No Problems | 14 | 13 | 4 | 10
  Anxiety/Depression: Week 18: Slight Problems | 9 | 6 | 5 | 2
  Anxiety/Depression: Week 18: Moderate Problems | 4 | 5 | 1 | 3
  Anxiety/Depression: Week 18: Severe Problems | 2 | 0 | 0 | 0
  Anxiety/Depression: Week 18: Extreme Problems | 0 | 0 | 0 | 0
  Anxiety/Depression: Week 21: number analyzed (Participants) | 24 | 24 | 13 | 12
  Anxiety/Depression: Week 21: No Problems | 12 | 12 | 8 | 2
  Anxiety/Depression: Week 21: Slight Problems | 7 | 4 | 4 | 6
  Anxiety/Depression: Week 21: Moderate Problems | 4 | 7 | 1 | 4
  Anxiety/Depression: Week 21: Severe Problems | 0 | 1 | 0 | 0
  Anxiety/Depression: Week 21: Extreme Problems | 1 | 0 | 0 | 0
  Anxiety/Depression: Week 24: number analyzed (Participants) | 21 | 18 | 13 | 8
  Anxiety/Depression: Week 24: No Problems | 10 | 10 | 8 | 3
  Anxiety/Depression: Week 24: Slight Problems | 8 | 3 | 5 | 2
  Anxiety/Depression: Week 24: Moderate Problems | 2 | 4 | 0 | 3
  Anxiety/Depression: Week 24: Severe Problems | 1 | 1 | 0 | 0
  Anxiety/Depression: Week 24: Extreme Problems | 0 | 0 | 0 | 0
  Anxiety/Depression: Week 27: number analyzed (Participants) | 15 | 14 | 6 | 5
  Anxiety/Depression: Week 27: No Problems | 7 | 7 | 4 | 1
  Anxiety/Depression: Week 27: Slight Problems | 4 | 4 | 2 | 1
  Anxiety/Depression: Week 27: Moderate Problems | 3 | 1 | 0 | 3
  Anxiety/Depression: Week 27: Severe Problems | 1 | 2 | 0 | 0
  Anxiety/Depression: Week 27: Extreme Problems | 0 | 0 | 0 | 0
  Anxiety/Depression: Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Anxiety/Depression: Week 90: No Problems | 1 |  |  |
  Anxiety/Depression: Week 90: Slight Problems | 0 |  |  |
  Anxiety/Depression: Week 90: Moderate Problems | 0 |  |  |
  Anxiety/Depression: Week 90: Severe Problems | 0 |  |  |
  Anxiety/Depression: Week 90: Extreme Problems | 0 |  |  |

15. Secondary Outcome: Phase 2 Cohorts: Change From Baseline in the EuroQol Visual Analogue Scale (EQ-VAS) Score
Description: The EQ-VAS recorded the participant's self-rated health on a vertical VAS, where the end points were labeled "the best health you can imagine" and "the worst health you can imagine." The EQ-VAS could be used as a quantitative measure of a health outcome that reflected the participant's own judgment. The EQ-VAS recorded the participant's self-rated health on a vertical VAS, with a score numbered from 0 to 100, where '100 meant the best health you can imagine' and '0 meant the worst health you can imagine".
Time Frame: Baseline, Week 3, Week 6, Week 9, Week 12, Week 15, Week 18, Week 21, Week 24, Week 27 and Week 90
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum+5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum+5-FU | Phase 2 Cohort 3: Magrolimab + Docetaxel
Number analyzed (Participants) | 52 | 52 | 32 | 41
score on scale
  Baseline: number analyzed (Participants) | 52 | 50 | 27 | 36
  Baseline | 61.9 (20.96) | 64.0 (23.15) | 59.8 (24.86) | 62.0 (22.21)
  Change at Week 3: number analyzed (Participants) | 41 | 42 | 23 | 27
  Change at Week 3 | -3.7 (20.80) | 4.3 (20.72) | 4.1 (17.88) | -0.3 (16.20)
  Change at Week 6: number analyzed (Participants) | 30 | 38 | 14 | 26
  Change at Week 6 | 2.2 (14.82) | 5.7 (24.75) | 1.1 (15.71) | -2.1 (16.37)
  Change at Week 9: number analyzed (Participants) | 29 | 29 | 16 | 20
  Change at Week 9 | -1.0 (18.19) | 2.5 (16.89) | 6.6 (18.50) | 4.4 (20.74)
  Change at Week 12: number analyzed (Participants) | 31 | 32 | 16 | 18
  Change at Week 12 | 4.5 (18.65) | 7.9 (23.02) | 5.9 (19.60) | -4.5 (14.55)
  Change at Week 15: number analyzed (Participants) | 31 | 29 | 11 | 18
  Change at Week 15 | 0.1 (18.79) | 10.5 (23.60) | 3.2 (15.05) | -1.1 (12.86)
  Change at Week 18: number analyzed (Participants) | 29 | 25 | 11 | 15
  Change at Week 18 | -1.2 (19.34) | 7.4 (23.33) | 3.8 (20.11) | -8.1 (17.77)
  Change at Week 21: number analyzed (Participants) | 24 | 24 | 11 | 11
  Change at Week 21 | 0.5 (18.59) | 1.1 (21.12) | 4.0 (20.15) | -8.5 (16.71)
  Change at Week 24: number analyzed (Participants) | 21 | 17 | 12 | 7
  Change at Week 24 | 0.2 (22.05) | 6.0 (22.45) | 2.1 (20.72) | -13.9 (19.17)
  Change at Week 27: number analyzed (Participants) | 14 | 13 | 6 | 5
  Change at Week 27 | -10.0 (19.32) | -0.9 (22.46) | 10.0 (21.45) | -9.0 (23.56)
  Change at Week 90: number analyzed (Participants) | 1 | 0 | 0 | 0
  Change at Week 90 | 25.0 (NA) — Standard Deviation can not be estimated for one participant. |  |  |

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 129 weeks; Adverse Events: Up to 73 weeks plus 30 days
Description: All-cause mortality: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Arm/Group | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU | Safety Run-in Cohort 2: Magrolimab + Docetaxel | Phase 2 Cohort 3: Magrolimab + Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/6 | 25/52 | 22/54 | 9/32 | 6/8 | 24/41
Serious Adverse Events (participants affected / at risk) | 4/6 | 26/52 | 24/53 | 15/29 | 6/7 | 24/41
Other Adverse Events (participants affected / at risk) | 6/6 | 49/52 | 53/53 | 28/29 | 7/7 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU (N=6) | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU (N=52) | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU (N=53) | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU (N=29) | Safety Run-in Cohort 2: Magrolimab + Docetaxel (N=7) | Phase 2 Cohort 3: Magrolimab + Docetaxel (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 1 | 3 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral cavity fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 2 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 2 | 3 | 1 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tongue abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Stoma site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Middle cerebral artery stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 1 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Septic shock from neutropenic colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1: Magrolimab + Pembrolizumab + Platinum + 5-FU (N=6) | Phase 2 Cohort 1 Arm A: Magrolimab + Pembrolizumab + Platinum + 5-FU (N=52) | Phase 2 Cohort 1 Arm B: Pembrolizumab + Platinum + 5-FU (N=53) | Phase 2 Cohort 1 Arm C: Magrolimab + Zimberelimab + Platinum + 5-FU (N=29) | Safety Run-in Cohort 2: Magrolimab + Docetaxel (N=7) | Phase 2 Cohort 3: Magrolimab + Docetaxel (N=41)
Anaemia (Blood and lymphatic system disorders) | 5 | 43 | 37 | 21 | 5 | 28
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 7 | 4 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 9 | 6 | 2 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 16 | 12 | 7 | 1 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 16 | 20 | 5 | 0 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 2 | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 6 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 3 | 4 | 1 | 0 | 2
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 18 | 16 | 4 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 11 | 13 | 7 | 2 | 14
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 3 | 3 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 5 | 1 | 0 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 5 | 1 | 0 | 3
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 19 | 23 | 11 | 2 | 15
Oral dysaesthesia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 5 | 7 | 18 | 9 | 2 | 10
Vomiting (Gastrointestinal disorders) | 1 | 6 | 7 | 7 | 0 | 6
Asthenia (General disorders) | 1 | 16 | 15 | 10 | 0 | 7
Chills (General disorders) | 1 | 3 | 1 | 3 | 1 | 1
Fatigue (General disorders) | 5 | 12 | 11 | 9 | 4 | 14
Influenza like illness (General disorders) | 1 | 1 | 1 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 5 | 4 | 3 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 3 | 0 | 2 | 1 | 5
Pain (General disorders) | 0 | 4 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 6 | 3 | 3 | 1 | 5
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 2
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 2 | 4 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 4 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 2 | 3 | 1 | 0 | 2
Stoma site infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 6 | 1 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5 | 5 | 3 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 5 | 3 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 7 | 2 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 2 | 2 | 4 | 0 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 3 | 4 | 2 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 3 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2 | 3 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 6 | 0 | 2 | 0 | 4
Neutrophil count decreased (Investigations) | 2 | 11 | 2 | 4 | 4 | 9
Platelet count decreased (Investigations) | 5 | 8 | 8 | 8 | 3 | 1
Weight decreased (Investigations) | 0 | 3 | 7 | 5 | 2 | 2
White blood cell count decreased (Investigations) | 4 | 11 | 4 | 4 | 2 | 8
Decreased appetite (Metabolism and nutrition disorders) | 3 | 14 | 10 | 3 | 3 | 10
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 0 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 4 | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 7 | 10 | 6 | 0 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 10 | 8 | 8 | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 7 | 9 | 8 | 1 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 6 | 2 | 8 | 0 | 5
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 4 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 4 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 5 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 1 | 3 | 2 | 2
Headache (Nervous system disorders) | 1 | 10 | 5 | 8 | 2 | 7
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 3
Presyncope (Nervous system disorders) | 1 | 3 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 5 | 4 | 3 | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7 | 5 | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 6 | 5 | 1 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 3 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 4 | 3 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 3 | 3 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04854499/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT04854499/SAP_001.pdf